CLINICAL TRIAL: NCT01025336
Title: A Study To Evaluate The Persistence Of The Antibody Response Elicited By 13-Valent Pneumococcal Conjugate Vaccine (13vPnC) In Healthy Adults Who Have Previously Been Vaccinated With Either 2 Doses Of 13vPnC Or 13vPnC And 23-Valent Pneumococcal Polysaccharide Vaccine In Different Sequential Order In Study 6115A1-3010 Or 6115A1 3005
Brief Title: Study Evaluating Persistence Of Antibody Response Elicited By 13vPnC In Healthy Adults Previously Vaccinated
Acronym: AB PERSISTENCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 6115A1-3018; B1851029
Record Dates: First submitted 2009-11-20; First posted 2009-12-03 (Estimated); Results first posted 2012-06-20 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: Antibody persistence
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 23vPS Naive (Other): Group 1.1 13vPnC/13vPnC Group 1.2 13vPnC/23vPS Group 2 23vPS/13vPNC
  Interventions: Other: Blood draw
- Prior 23vPS>/= 5 years (Other): Group 1 13vPnC/13vPnC Group 2 23vPS/13vPnC
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — Group 1.1- 0.5 mL dose of 13vPnC was administered in the deltoid muscle at year 0 and 0.5 mL dose of 13vPnC was administered in the deltoid muscle at year 1 Group 1.2- 0.5 mL dose of 13vPnC was administered in the deltoid muscle at year 0 and 0.5 mL dose of 23vPS was administered in the deltoid muscle at year 1 Group 2- 0.5 mL dose of 23vPS was administered in the deltoid muscle at year 0 and 0.5 mL dose of 13vPnC was administered in the deltoid muscle at year 1
  Arms: 23vPS Naive
Other: Blood draw — Group 1- 0.5 mL dose of 13vPnC was administered in the deltoid muscle at year 0 and year 1 Group 2- 0.5 mL dose of 23vPS was administered in the deltoid muscle at year 0 and 0.5 mL dose of 13vPNC was administered in the deltoid muscle at year 1
  Arms: Prior 23vPS>/= 5 years

SUMMARY:
The purpose of this study is to evaluate the levels of antibodies 1 year after receiving the second vaccine dose in two groups of adults over the age of 60: (1) those who have previously received 2 doses of 13-valent pneumococcal conjugate vaccine (13vPnC) and (2) those who have previously received 1 dose of 13vPnc and 1 dose of 23-valent pneumococcal polysaccharide vaccine (23vPS). This study will also assess whether the use of the 2 vaccines, 13vPnC and 23vPS, administered in different sequential order results in different prolonged antibody levels. This study is limited to individuals who participated in either study 6115A1-3010 (NCT00574548) or 6115A1-3005 (NCT00546572).

ELIGIBILITY:
Inclusion Criteria:

* Only study volunteers who received both assigned vaccinations at visit 1 and visit 4 when they participated in either study 6115A1-3010 (NCT00574548) or 6115A1-3005 (NCT00546572)

Exclusion Criteria:

* Vaccination with any licensed or experimental pneumococcal vaccine since being enrolled in the 6115A1-3005 (NCT00546572) or 6115A1-3010 (NCT00574548) study (other than study vaccines permitted in 6115A1-3010 or 6115A1-3005)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 962 (Actual)
Dates: Start 2009-12; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (28):
- United States (28):
  - Pfizer Investigational Site, Chandler, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Pinellas Park, Florida
  - Pfizer Investigational Site, Meridian, Idaho
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Cary, North Carolina
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Corvallis, Oregon
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Carnegie, Pennsylvania
  - Pfizer Investigational Site, Grove City, Pennsylvania
  - Pfizer Investigational Site, Jefferson, Pennsylvania
  - Pfizer Investigational Site, Penndel, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, Mt. Pleasant, South Carolina
  - Pfizer Investigational Site, Bristol, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Seattle, Washington

REFERENCES:
- [Derived] Schmoele-Thoma B, van Cleeff M, Greenberg RN, Gurtman A, Jones TR, Sundaraiyer V, Gruber WC, Scott DA. Persistence of antibodies 1 year after sequential administration of the 13-valent pneumococcal conjugate vaccine and the 23-valent pneumococcal polysaccharide vaccine in adults. Hum Vaccin Immunother. 2019;15(3):575-583. doi: 10.1080/21645515.2018.1538618. Epub 2019 Jan 16. PMID 30648932
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6115A1-3018&StudyName=Study%20Evaluating%20Persistence%20Of%20Antibody%20Response%20Elicited%20By%2013vPnC%20In%20Healthy%20Adults%20%20Previously%20Vaccinated

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only participants who completed Parent Study 6115A1-3010 (NCT00574548) or Parent Study 6115A1-3005 (NCT00546572) were enrolled in this follow-up study 6115A1-3018 (NCT01025336).
Groups:
- 13vPnC/13vPnC Group (23vPS Naïve): Participants aged 60 to 64 years old who had never received 23-valent pneumococcal polysaccharide vaccine (23vPS) prior to enrollment into the parent study (NCT00574548), completed study NCT00574548 receiving 13 valent pneumococcal conjugate (13vPnC) administered as a single dose 0.5 milliliter (mL) intramuscularly (IM) at Year 0 (Vaccination 1) and at Year 1 (Vaccination 2)
- 13vPnC/23vPS Group (23vPS Naïve): Participants aged 60 to 64 years old who had never received 23vPS prior to enrollment into the parent study (NCT00574548), completed study NCT00574548 receiving 13vPnC administered as a single dose 0.5 mL IM at Year 0 (Vaccination 1) and 23vPS administered as a single dose 0.5 mL IM at Year 1 (Vaccination 2)
- 23vPS/13vPnC Group (23vPS Naïve): Participants aged 60 to 64 years old who had never been vaccinated with 23vPS prior to enrollment into the parent study (NCT00574548), who completed study NCT00574548 receiving 23vPS administered as a single dose 0.5 mL IM at Year 0 (Vaccination 1) and 13vPnC administered as a single dose 0.5 mL IM at Year 1 (Vaccination 2)
- 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior): Participants aged 70 years of age or greater previously vaccinated with 23vPS greater than or equal to (≥) 5 years before enrollment in the parent study (NCT00546572), who completed study NCT00546572 receiving 13vPnC administered as a single dose 0.5 mL IM at Year 0 (Vaccination 1) and at Year 1 (Vaccination 2)
- 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior): Participants aged 70 years of age or greater previously vaccinated with 23vPS ≥5 years before enrollment in the parent study (NCT00546572), who completed study NCT00546572 receiving 23vPS administered as a single dose 0.5 mL IM at Year 0 (Vaccination 1) and 13vPnC administered as a single dose 0.5 mL IM at Year 1 (Vaccination 2)
Period: Overall Study
Arm/Group | 13vPnC/13vPnC Group (23vPS Naïve) | 13vPnC/23vPS Group (23vPS Naïve) | 23vPS/13vPnC Group (23vPS Naïve) | 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) | 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior)
Started | 130 | 210 | 179 | 221 | 222
Completed | 130 | 210 | 179 | 219 | 222
Not Completed | 0 | 0 | 0 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC/13vPnC Group (23vPS Naïve) | 13vPnC/23vPS Group (23vPS Naïve) | 23vPS/13vPnC Group (23vPS Naïve) | 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) | 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior) | Total
Number analyzed (Participants) | 130 | 210 | 179 | 221 | 222 | 962
Age Continuous [Mean (Standard Deviation); unit: Years] | 64.0 (1.4) | 64.1 (1.4) | 64.2 (1.4) | 78.3 (4.5) | 77.8 (4.1) | 70.5 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 125 | 102 | 114 | 115 | 532
  Male | 54 | 85 | 77 | 107 | 107 | 430

OUTCOME MEASURES:

1. Primary Outcome: Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titer (GMT) Antibody Persistence 1 Year After Vaccination (Vax) 2 in Parent Study 6115A1-3010 (NCT00574548)
Description: Antibody GMTs as measured by OPA assay for 13 pneumococcal serotypes (serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F). Confidence intervals (CIs) for the GMTs are back transformations of a confidence interval based on the Student t distribution for the mean logarithm of the titers.
Time Frame: Month 1/Year 2 (Baseline) (Follow-up Study 6115A1-3018; NCT01025336)
Population: All-Available Immunogenicity Population included all participants enrolled in 6115A1-3018 (NCT01025336) with a valid and determinate assay result who received both vaccinations in either parent study 6115A1-3010 (NCT00574548) or 6115A1-3005 (NCT00546572). N=number of participants with valid and determinate antibody titer for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- 13vPnC/13vPnC Group (23vPs Naïve): Participants aged 60 to 64 years old who had never received 23-valent pneumococcal polysaccharide vaccine (23vPS) prior to enrollment into the parent study 6115A1-3010 (NCT00574548), completed study NCT00574548 receiving 13 valent pneumococcal conjugate (13vPnC) administered as a single dose 0.5 milliliter (mL) intramuscularly (IM) at Year 0 (Vaccination 1) and at Year 1 (Vaccination 2)
- 13vPnC/23vPS Group (23vPS Naïve): Participants aged 60 to 64 years old who had never received 23vPS prior to enrollment into the parent study 6115A-3010 6115A1-3010(NCT00574548), completed study NCT00574548 receiving 13vPnC administered as a single dose 0.5 mL IM at Year 0 (Vaccination 1) and 23vPS administered as a single dose 0.5 mL IM at Year 1 (Vaccination 2)
- 23vPS/13vPnC Group (23vPS Naïve): Participants aged 60 to 64 years old who had never been vaccinated with 23vPS prior to enrollment into the parent study 6115A1-3010 (NCT00574548), who completed study NCT00574548 receiving 23vPS administered as a single dose 0.5 mL IM at Year 0 (Vaccination 1) and 13vPnC administered as a single dose 0.5 mL IM at Year 1 (Vaccination 2)
Arm/Group | 13vPnC/13vPnC Group (23vPs Naïve) | 13vPnC/23vPS Group (23vPS Naïve) | 23vPS/13vPnC Group (23vPS Naïve)
Number analyzed (Participants) | 129 | 209 | 179
titer
  Serotype 1 | 54 [40.8 to 71.0] | 52 [40.9 to 65.5] | 36 [27.1 to 46.7]
  Serotype 3 | 19 [15.0 to 23.5] | 27 [22.2 to 32.3] | 18 [14.4 to 21.9]
  Serotype 4 | 328 [229.0 to 469.0] | 355 [264.7 to 475.9] | 183 [127.7 to 263.2]
  Serotype 5 | 29 [20.4 to 41.4] | 76 [58.0 to 99.7] | 44 [32.9 to 59.6]
  Serotype 6A | 316 [216.5 to 461.2] | 225 [163.6 to 308.3] | 102 [71.4 to 146.9]
  Serotype 6B | 785 [540.6 to 1140.2] | 593 [441.4 to 797.3] | 324 [225.0 to 466.1]
  Serotype 7F | 247 [160.4 to 380.9] | 412 [313.1 to 541.2] | 145 [100.3 to 210.7]
  Serotype 9V | 211 [134.3 to 330.9] | 221 [154.2 to 316.0] | 129 [84.5 to 196.5]
  Serotype 14 | 379 [273.6 to 526.2] | 416 [316.2 to 548.2] | 383 [286.9 to 510.6]
  Serotype 18C | 393 [271.3 to 569.3] | 527 [401.7 to 690.5] | 337 [240.7 to 471.7]
  Serotype 19A | 244 [189.1 to 314.1] | 313 [263.1 to 372.3] | 170 [134.4 to 214.8]
  Serotype 19F | 256 [182.4 to 359.0] | 426 [343.7 to 527.7] | 195 [145.1 to 262.1]
  Serotype 23F | 110 [73.9 to 165.0] | 64 [47.6 to 86.5] | 35 [25.6 to 48.6]

2. Secondary Outcome: Serotype-Specific Pneumococcal OPA GMT Antibody Persistence 1 Year After Vaccination 2 Relative to 1 Month After Vaccination 2 (Parent Study 6115A1-3010; NCT00574548)
Description: Antibody GMTs as measured by OPA assay for 13 pneumococcal serotypes (serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F). CI for the GMTs are back transformations of a CI based on the Student t distribution for the mean logarithm of the concentrations.
Time Frame: Month 1/Year 1 (Parent study/NCT00574548), Month 1/Year 2 (Follow-up Study/NCT01025336)
Population: All-Available Immunogenicity Population; N=number of participants with valid and determinate assay result for specified serotype at both 1 Month Postvaccination 2 and 1 Year Postvaccination 2 blood draws.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- 13vPnC/13vPnC Group (23vPS Naïve): Participants aged 60 to 64 years old who had never received 23vPS prior to enrollment into the parent study 6115A1-3010 (NCT00574548), completed study NCT00574548 receiving 13vPnC administered as a single dose 0.5 mL IM at Year 0 (Vaccination 1) and at Year 1 (Vaccination 2)
- 13vPnC/23vPS Group (23vPS Naïve): Participants aged 60 to 64 years old who had never received 23vPS prior to enrollment into the parent study 6115A1-3010 (NCT00574548), completed study NCT00574548 receiving 13vPnC administered as a single dose 0.5 mL IM at Year 0 (Vaccination 1) and 23vPS administered as a single dose 0.5 mL IM at Year 1 (Vaccination 2)
Arm/Group | 13vPnC/13vPnC Group (23vPS Naïve) | 13vPnC/23vPS Group (23vPS Naïve) | 23vPS/13vPnC Group (23vPS Naïve)
Number analyzed (Participants) | 126 | 204 | 175
titer
  Serotype 1, 1 Month Post Vax 2 | 141 [110.4 to 179.7] | 149 [123.5 to 180.6] | 70 [53.4 to 91.2]
  Serotype 1, 1 Year Post Vax 2 | 54 [40.7 to 70.4] | 52 [41.1 to 66.1] | 36 [27.6 to 47.9]
  Serotype 3, 1 Month Post Vax 2 | 87 [73.7 to 103.8] | 130 [112.8 to 150.3] | 50 [40.2 to 63.1]
  Serotype 3, 1 Year Post Vax 2 | 18 [14.6 to 22.9] | 27 [22.2 to 32.5] | 18 [14.5 to 22.2]
  Serotype 4, 1 Month Post Vax 2 | 1284 [992.3 to 1661.9] | 1375 [1137.0 to 1663.8] | 898 [684.1 to 1179.5]
  Serotype 4, 1 Year Post Vax 2 | 318 [220.9 to 458.7] | 369 [276.1 to 493.9] | 203 [142.0 to 291.4]
  Serotype 5, 1 Month Post Vax 2 | 95 [67.1 to 133.2] | 223 [180.7 to 276.3] | 80 [59.7 to 108.3]
  Serotype 5, 1 Year Post Vax 2 | 29 [20.3 to 42.5] | 72 [54.6 to 95.1] | 41 [30.3 to 56.2]
  Serotype 6A, 1 Month Post Vax 2 | 2120 [1614.1 to 2783.9] | 1307 [1021.4 to 1672.8] | 933 [682.1 to 1276.2]
  Serotype 6A, 1 Year Post Vax 2 | 304 [207.7 to 446.3] | 266 [195.2 to 362.6] | 115 [79.3 to 166.3]
  Serotype 6B, 1 Month Post Vax 2 | 1683 [1253.6 to 2258.3] | 1232 [965.9 to 1570.4] | 740 [534.8 to 1024.2]
  Serotype 6B, 1 Year Post Vax 2 | 847 [590.8 to 1214.8] | 637 [476.3 to 851.6] | 352 [244.8 to 505.5]
  Serotype 7F, 1 Month Post Vax 2 | 306 [201.8 to 462.5] | 667 [531.5 to 836.8] | 131 [87.8 to 496.9]
  Serotype 7F, 1 Year Post Vax 2 | 237 [152.2 to 369.9] | 412 [313.2 to 541.5] | 148 [101.4 to 215.1]
  Serotype 9V, 1 Month Post Vax 2 | 385 [252.6 to 586.8] | 419 [298.6 to 588.0] | 122 [80.0 to 186.1]
  Serotype 9V, 1 Year Post Vax 2 | 221 [139.8 to 350.8] | 224 [155.9 to 321.6] | 139 [90.6 to 213.1]
  Serotype 14, 1 Month Post Vax 2 | 434 [311.6 to 605.6] | 639 [487.8 to 836.3] | 426 [312.7 to 580.5]
  Serotype 14, 1 Year Post Vax 2 | 380 [273.4 to 528.8] | 406 [306.7 to 537.0] | 388 [290.7 to 517.2]
  Serotype 18C, 1 Month Post Vax 2 | 972 [732.4 to 1290.1] | 1092 [879.6 to 1356.2] | 549 [395.9 to 761.1]
  Serotype 18C, 1 Year Post Vax 2 | 373 [255.6 to 544.2] | 513 [389.6 to 676.7] | 331 [235.3 to 467.0]
  Serotype 19A, 1 Month Post Vax 2 | 365 [295.0 to 450.7] | 513 [445.6 to 590.5] | 282 [230.3 to 344.4]
  Serotype 19A, 1 Year Post Vax 2 | 213 [163.6 to 276.3] | 295 [246.6 to 352.7] | 167 [132.0 to 210.5]
  Serotype 19F, 1 Month Post Vax 2 | 493 [365.0 to 664.7] | 835 [685.5 to 1015.9] | 264 [196.3 to 355.8]
  Serotype 19F, 1 Year Post Vax 2 | 255 [180.5 to 360.8] | 425 [340.9 to 529.2] | 197 [146.4 to 266.2]
  Serotype 23F, 1 Month Post Vax 2 | 543 [392.9 to 749.4] | 218 [164.8 to 288.0] | 109 [76.4 to 156.2]
  Serotype 23F, 1 Year Post Vax 2 | 108 [71.9 to 162.3] | 63 [46.4 to 84.5] | 38 [27.1 to 52.2]
Statistical Analysis 1: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 1: Geometric mean fold rise (GMFR) was calculated using all participants with available data from both the 1 Month Postvaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.4, 95% CI 2-sided [0.32 to 0.46] — CIs for the GMFR are back transformations of a CI based on the Student t distribution for the mean logarithm of the concentrations
Statistical Analysis 2: Comparison: 13vPnC/23vPS Group (23vPS Naïve); Serotype 1: GMFR was calculated using all participants with available data from both the 1 Month Postvaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.3, 95% CI 2-sided [0.30 to 0.41] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; geometric mean fold rise = 0.5, 95% CI 2-sided [0.44 to 0.61] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 3: GMFR was calculated using all participants with available data from both the 1 Month Postvaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.2, 95% CI 2-sided [0.17 to 0.25] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; geometric mean fold rise = 0.2, 95% CI 2-sided [0.18 to 0.24] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; geometric mean fold rise = 0.4, 95% CI 2-sided [0.31 to 0.41] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 4: GMFR was calculated using all participants with available data from both the 1 Month Postvaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.2, 95% CI 2-sided [0.19 to 0.32] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; geometric mean fold rise = 0.3, 95% CI 2-sided [0.22 to 0.33] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; geometric mean fold rise = 0.2, 95% CI 2-sided [0.17 to 0.30] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 5: GMFR was calculated using all participants with available data from both the 1 Month Postvaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.3, 95% CI 2-sided [0.25 to 0.39] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 2, analysis 10]; Test type: Superiority or Other; geometric mean fold rise = 0.3, 95% CI 2-sided [0.27 to 0.38] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 2, analysis 10]; Test type: Superiority or Other; geometric mean fold rise = 0.5, 95% CI 2-sided [0.44 to 0.60] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 6A: GMFR was calculated using all participants with available data from both the 1 Month Postvaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.1, 95% CI 2-sided [0.10 to 0.20] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 14: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; geometric mean fold rise = 0.2, 95% CI 2-sided [0.17 to 0.25] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 15: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; geometric mean fold rise = 0.1, 95% CI 2-sided [0.09 to 0.16] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 16: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 6B: GMFR was calculated using all participants with available data from both the 1 Month Postvaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.5, 95% CI 2-sided [0.41 to 0.62] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 17: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 2, analysis 16]; Test type: Superiority or Other; geometric mean fold rise = 0.5, 95% CI 2-sided [0.43 to 0.62] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 18: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 2, analysis 16]; Test type: Superiority or Other; geometric mean fold rise = 0.5, 95% CI 2-sided [0.38 to 0.59] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 19: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 7F: GMFR was calculated using all participants with available data from both the 1 Month Postvaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.8, 95% CI 2-sided [0.60 to 1.00] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 20: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 2, analysis 19]; Test type: Superiority or Other; geometric mean fold rise = 0.6, 95% CI 2-sided [0.51 to 0.75] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 21: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 2, analysis 19]; Test type: Superiority or Other; geometric mean fold rise = 1.1, 95% CI 2-sided [0.86 to 1.46] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 22: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 9V: GMFR was calculated using all participants with available data from both the 1 Month Postvaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.6, 95% CI 2-sided [0.41 to 0.80] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 23: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 2, analysis 22]; Test type: Superiority or Other; geometric mean fold rise = 0.5, 95% CI 2-sided [0.39 to 0.73] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 24: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 2, analysis 22]; Test type: Superiority or Other; geometric mean fold rise = 1.1, 95% CI 2-sided [0.78 to 1.67] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 25: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 14: GMFR was calculated using all participants with available data from both the 1 Month Postvaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.9, 95% CI 2-sided [0.71 to 1.08] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 26: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 2, analysis 25]; Test type: Superiority or Other; geometric mean fold rise = 0.6, 95% CI 2-sided [0.54 to 0.75] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 27: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 2, analysis 25]; Test type: Superiority or Other; geometric mean fold rise = 0.9, 95% CI 2-sided [0.78 to 1.06] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 28: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 18C: GMFR was calculated using all participants with available data from both the 1 Month Postvaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.4, 95% CI 2-sided [0.29 to 0.51] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 29: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 2, analysis 28]; Test type: Superiority or Other; geometric mean fold rise = 0.5, 95% CI 2-sided [0.39 to 0.56] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 30: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 2, analysis 28]; Test type: Superiority or Other; geometric mean fold rise = 0.6, 95% CI 2-sided [0.53 to 0.69] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 31: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 19A: GMFR was calculated using all participants with available data from both the 1 Month Postvaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.6, 95% CI 2-sided [0.49 to 0.69] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 32: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 2, analysis 31]; Test type: Superiority or Other; geometric mean fold rise = 0.6, 95% CI 2-sided [0.52 to 0.63] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 33: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 2, analysis 31]; Test type: Superiority or Other; geometric mean fold rise = 0.6, 95% CI 2-sided [0.53 to 0.66] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 34: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 19F: GMFR was calculated using all participants with available data from both the 1 Month Postvaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.5, 95% CI 2-sided [0.42 to 0.64] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 35: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 2, analysis 34]; Test type: Superiority or Other; geometric mean fold rise = 0.5, 95% CI 2-sided [0.44 to 0.60] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 36: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 2, analysis 34]; Test type: Superiority or Other; geometric mean fold rise = 0.7, 95% CI 2-sided [0.63 to 0.88] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 37: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 23F: GMFR was calculated using all participants with available data from both the 1 Month Postvaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.2, 95% CI 2-sided [0.15 to 0.26] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 38: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 2, analysis 37]; Test type: Superiority or Other; geometric mean fold rise = 0.3, 95% CI 2-sided [0.23 to 0.35] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 39: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 2, analysis 37]; Test type: Superiority or Other; geometric mean fold rise = 0.3, 95% CI 2-sided [0.28 to 0.43] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Serotype-Specific Pneumococcal OPA GMT Antibody Persistence 1 Year After Vaccination 2 Relative to 1 Month After Vaccination 2 (Parent Study 6115A1-3005; NCT00546572)
Description: as for outcome 2
Time Frame: Month 1/Year 1 (Parent study/NCT00546572), Month 1/Year 2 (Follow-up Study/NCT01025336)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior): Participants at least 70 years of age or greater previously vaccinated with 23vPS ≥5 years before enrollment in the parent study 6115A1-3005 (NCT00546572), who completed study NCT00546572 receiving 13vPnC administered as a single dose 0.5 mL IM at Year 0 (Vaccination 1)and at Year 1 (Vaccination 2)
- 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior): Participants at least 70 years of age or greater previously vaccinated with 23vPS ≥5 years before enrollment in the parent study 6115A1-3005 (NCT00546572), who completed study NCT00546572 receiving 23vPS administered as a single dose 0.5 mL IM at Year 0 (Vaccination 1) and 13vPnC administered as a single dose 0.5 mL IM at Year 1 (Vaccination 2)
Arm/Group | 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) | 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior)
Number analyzed (Participants) | 216 | 217
titer
  Serotype 1, 1 Month Post Vax 2 | 80 [65.0 to 97.7] | 34 [27.2 to 43.7]
  Serotype 1, 1 Year Post Vax 2 | 39 [31.1 to 48.2] | 22 [17.4 to 27.6]
  Serotype 3, 1 Month Post Vax 2 | 50 [42.1 to 59.2] | 32 [26.1 to 38.9]
  Serotype 3, 1 Year Post Vax 2 | 20 [16.5 to 23.6] | 16 [13.2 to 19.1]
  Serotype 4, 1 Month Post Vax 2 | 437 [332.0 to 576.3] | 237 [173.5 to 325.1]
  Serotype 4, 1 Year Post Vax 2 | 311 [238.1 to 407.1] | 186 [138.3 to 250.2]
  Serotype 5, 1 Month Post Vax 2 | 62 [48.1 to 79.4] | 49 [37.4 to 63.7]
  Serotype 5, 1 Year Post Vax 2 | 58 [45.0 to 74.4] | 42 [31.7 to 54.8]
  Serotype 6A, 1 Month Post Vax 2 | 1088 [843.2 to 1404.7] | 569 [421.8 to 768.5]
  Serotype 6A, 1 Year Post Vax 2 | 257 [192.4 to 342.9] | 133 [97.4 to 182.1]
  Serotype 6B, 1 Month Post Vax 2 | 1516 [1173.7 to 1957.5] | 781 [574.8 to 1061.9]
  Serotype 6B, 1 Year Post Vax 2 | 561 [421.4 to 746.9] | 381 [282.6 to 514.5]
  Serotype 7F, 1 Month Post Vax 2 | 233 [166.5 to 324.8] | 135 [93.2 to 194.5]
  Serotype 7F, 1 Year Post Vax 2 | 173 [125.9 to 239.1] | 117 [82.8 to 165.4]
  Serotype 9V, 1 Month Post Vax 2 | 166 [113.8 to 241.5] | 91 [62.0 to 133.3]
  Serotype 9V, 1 Year Post Vax 2 | 83 [56.2 to 121.9] | 73 [49.9 to 105.9]
  Serotype 14, 1 Month Post Vax 2 | 216 [163.8 to 284.3] | 199 [146.9 to 270.8]
  Serotype 14, 1 Year Post Vax 2 | 209 [159.5 to 272.9] | 244 [184.5 to 321.9]
  Serotype 18C, 1 Month Post Vax 2 | 1015 [832.6 to 1237.6] | 523 [395.1 to 693.5]
  Serotype 18C, 1 Year Post Vax 2 | 553 [446.5 to 685.6] | 366 [277.2 to 482.9]
  Serotype 19A, 1 Month Post Vax 2 | 356 [297.6 to 425.6] | 255 [207.8 to 313.7]
  Serotype 19A, 1 Year Post Vax 2 | 228 [189.1 to 276.1] | 182 [147.7 to 225.2]
  Serotype 19F, 1 Month Post Vax 2 | 349 [274.7 to 444.5] | 178 [134.1 to 235.0]
  Serotype 19F, 1 Year Post Vax 2 | 274 [214.2 to 350.8] | 158 [119.1 to 210.6]
  Serotype 23F, 1 Month Post Vax 2 | 324 [250.8 to 419.8] | 113 [82.4 to 154.8]
  Serotype 23F, 1 Year Post Vax 2 | 102 [77.0 to 135.0] | 46 [33.9 to 61.7]
Statistical Analysis 1: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); Serotype 1: Geometric mean fold rises (GMFRs) were calculated using all subjects with available data from both the 1 Month Postvaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 0.5, 95% CI 2-sided [0.42 to 0.56] — Confidence intervals (CIs) are back transformations of a confidence interval based on the Student t distribution for the mean logarithm of the concentrations
Statistical Analysis 2: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Geometric mean fold rise = 0.6, 95% CI 2-sided [0.56 to 0.72] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); Serotype 3: Geometric mean fold rises (GMFRs) were calculated using all subjects with available data from both the 1 Month Postvaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 0.4, 95% CI 2-sided [0.35 to 0.45] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; Geometric mean fold rise = 0.5, 95% CI 2-sided [0.44 to 0.57] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); Serotype 4: Geometric mean fold rises (GMFRs) were calculated using all subjects with available data from both the 1 Month Postvaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 0.7, 95% CI 2-sided [0.60 to 0.85] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; Geometric mean fold rise = 0.8, 95% CI 2-sided [0.63 to 0.97] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); Serotype 5: Geometric mean fold rises (GMFRs) were calculated using all subjects with available data from both the 1 Month Postvaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 0.9, 95% CI 2-sided [0.81 to 1.08] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 8: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 3, analysis 7]; Test type: Superiority or Other; Geometric mean fold rise = 0.9, 95% CI 2-sided [0.74 to 0.99] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); Serotype 6A: Geometric mean fold rises (GMFRs) were calculated using all subjects with available data from both the 1 Month Postvaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 0.2, 95% CI 2-sided [0.19 to 0.29] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 10: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 3, analysis 9]; Test type: Superiority or Other; Geometric mean fold rise = 0.2, 95% CI 2-sided [0.19 to 0.29] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); Serotype 6B: Geometric mean fold rises (GMFRs) were calculated using all subjects with available data from both the 1 Month Postvaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 0.4, 95% CI 2-sided [0.31 to 0.45] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 12: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 3, analysis 11]; Test type: Superiority or Other; Geometric mean fold rise = 0.5, 95% CI 2-sided [0.40 to 0.59] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); Serotype 7F: Geometric mean fold rises (GMFRs) were calculated using all subjects with available data from both the 1 Month Postvaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 0.7, 95% CI 2-sided [0.58 to 0.96] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 14: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 3, analysis 13]; Test type: Superiority or Other; Geometric mean fold rise = 0.9, 95% CI 2-sided [0.67 to 1.13] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 15: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); Serotype 9V: Geometric mean fold rises (GMFRs) were calculated using all subjects with available data from both the 1 Month Postvaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 0.5, 95% CI 2-sided [0.37 to 0.67] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 16: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 3, analysis 15]; Test type: Superiority or Other; Geometric mean fold rise = 0.8, 95% CI 2-sided [0.57 to 1.12] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 17: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); Serotype 14: Geometric mean fold rises (GMFRs) were calculated using all subjects with available data from both the 1 Month Postvaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 1.0, 95% CI 2-sided [0.85 to 1.09] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 18: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 3, analysis 17]; Test type: Superiority or Other; Geometric mean fold rise = 1.2, 95% CI 2-sided [1.04 to 1.43] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 19: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); Serotype 18C: Geometric mean fold rises (GMFRs) were calculated using all subjects with available data from both the 1 Month Postvaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 0.5, 95% CI 2-sided [0.48 to 0.62] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 20: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 3, analysis 19]; Test type: Superiority or Other; Geometric mean fold rise = 0.7, 95% CI 2-sided [0.59 to 0.83] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 21: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); Serotype 19A: Geometric mean fold rises (GMFRs) were calculated using all subjects with available data from both the 1 Month Postvaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 0.6, 95% CI 2-sided [0.57 to 0.72] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 22: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 3, analysis 21]; Test type: Superiority or Other; Geometric mean fold rise = 0.7, 95% CI 2-sided [0.65 to 0.79] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 23: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); Serotype 19F: Geometric mean fold rises (GMFRs) were calculated using all subjects with available data from both the 1 Month Postvaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 0.8, 95% CI 2-sided [0.66 to 0.93] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 24: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 3, analysis 23]; Test type: Superiority or Other; Geometric mean fold rise = 0.9, 95% CI 2-sided [0.75 to 1.05] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 25: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); Serotype 23F: Geometric mean fold rises (GMFRs) were calculated using all subjects with available data from both the 1 Month Postvaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 0.3, 95% CI 2-sided [0.27 to 0.37] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 26: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 3, analysis 25]; Test type: Superiority or Other; Geometric mean fold rise = 0.4, 95% CI 2-sided [0.34 to 0.48] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Serotype-Specific Pneumococcal OPA GMT Antibody Persistence 1 Year After Vaccination 2 Relative to Before Vaccination 2 (Parent Study 6115A1-3010; NCT00574548)
Description: as for outcome 2
Time Frame: Month 0/Year 1 (Parent Study NCT00574548), Month 1/Year 2 (Follow-up Study NCT01025336)
Population: All-Available Immunogenicity Population; N=number of participants with valid and determinate assay result for specified serotype at both the Prevaccination 2 and 1 Year Postvaccination 2 blood draws.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC/13vPnC Group (23vPS Naïve) | 13vPnC/23vPS Group (23vPS Naïve) | 23vPS/13vPnC Group (23vPS Naïve)
Number analyzed (Participants) | 124 | 204 | 173
titer
  Serotype 1, Pre Vax 2 | 52 [38.2 to 69.5] | 56 [44.4 to 70.6] | 44 [33.0 to 57.7]
  Serotype 1, 1 Year Post Vax 2 | 52 [39.6 to 69.0] | 50 [39.7 to 63.9] | 34 [26.2 to 45.1]
  Serotype 3, Pre Vax 2 | 19 [14.5 to 24.1] | 23 [18.6 to 28.1] | 26 [20.3 to 32.4]
  Serotype 3, 1 Year Post Vax 2 | 18 [14.2 to 22.3] | 26 [21.4 to 31.6] | 18 [14.7 to 22.4]
  Serotype 4, Pre Vax 2 | 710 [504.4 to 998.7] | 591 [437.9 to 798.0] | 350 [242.0 to 506.6]
  Serotype 4, 1 Year Post Vax 2 | 376 [264.2 to 534.0] | 414 [312.3 to 548.2] | 209 [144.6 to 302.1]
  Serotype 5, Pre Vax 2 | 39 [26.2 to 56.7] | 66 [48.9 to 87.8] | 49 [36.4 to 67.1]
  Serotype 5, 1 Year Post Vax 2 | 29 [20.4 to 42.1] | 73 [55.3 to 96.4] | 43 [31.9 to 58.2]
  Serotype 6A, Pre Vax 2 | 540 [347.1 to 838.8] | 656 [484.0 to 888.4] | 85 [56.3 to 127.7]
  Serotype 6A, 1 Year Post Vax 2 | 331 [227.1 to 483.3] | 251 [183.4 to 343.3] | 108 [74.7 to 157.3]
  Serotype 6B, Pre Vax 2 | 459 [292.2 to 719.9] | 430 [304.8 to 605.6] | 192 [128.4 to 286.0]
  Serotype 6B, 1 Year Post Vax 2 | 781 [529.8 to 1150.8] | 580 [427.9 to 786.8] | 298 [203.8 to 435.6]
  Serotype 7F, Pre Vax 2 | 146 [89.4 to 237.1] | 133 [92.4 to 191.0] | 71 [46.9 to 107.6]
  Serotype 7F, 1 Year Post Vax 2 | 244 [155.7 to 383.4] | 414 [313.8 to 546.5] | 146 [99.7 to 212.8]
  Serotype 9V, Pre Vax 2 | 96 [58.3 to 158.4] | 79 [53.2 to 116.2] | 50 [32.4 to 78.5]
  Serotype 9V, 1 Year Post Vax 2 | 201 [125.8 to 320.2] | 212 [147.4 to 306.4] | 147 [95.8 to 226.8]
  Serotype 14, Pre Vax 2 | 241 [159.6 to 364.0] | 290 [208.6 to 403.1] | 302 [214.2 to 425.3]
  Serotype 14, 1 Year Post Vax 2 | 383 [274.1 to 534.2] | 420 [317.0 to 556.1] | 367 [272.9 to 493.4]
  Serotype 18C, Pre Vax 2 | 403 [273.8 to 592.0] | 462 [346.1 to 615.8] | 339 [236.2 to 487.4]
  Serotype 18C, 1 Year Post Vax 2 | 398 [274.1 to 579.1] | 513 [389.5 to 676.1] | 349 [247.8 to 492.2]
  Serotype 19A, Pre Vax 2 | 203 [151.3 to 271.8] | 209 [170.3 to 257.6] | 153 [117.3 to 199.5]
  Serotype 19A, 1 Year Post Vax 2 | 253 [197.2 to 325.7] | 296 [248.3 to 353.0] | 169 [133.0 to 214.6]
  Serotype 19F, Pre Vax 2 | 114 [72.7 to 177.5] | 183 [135.0 to 247.7] | 127 [89.7 to 180.1]
  Serotype 19F, 1 Year Post Vax 2 | 238 [165.2 to 341.7] | 419 [334.2 to 524.2] | 190 [139.8 to 258.7]
  Serotype 23F, Pre Vax 2 | 90 [58.5 to 139.9] | 90 [65.4 to 123.6] | 30 [21.2 to 42.1]
  Serotype 23F, 1 Year Post Vax 2 | 104 [67.9 to 158.6] | 66 [48.7 to 88.9] | 36 [26.3 to 50.6]
Statistical Analysis 1: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 1: GMFR was calculated using all participants with available data from both the Prevaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 1.0, 95% CI 2-sided [0.85 to 1.22] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Geometric mean fold rise = 0.9, 95% CI 2-sided [0.79 to 1.02] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Geometric mean fold rise = 0.8, 95% CI 2-sided [0.69 to 0.90] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 3: GMFR was calculated using all participants with available data from both the Prevaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 1.0, 95% CI 2-sided [0.82 to 1.10] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; Geometric mean fold rise = 1.1, 95% CI 2-sided [0.98 to 1.32] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; Geometric mean fold rise = 0.7, 95% CI 2-sided [0.62 to 0.81] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 4: GMFR was calculated using all participants with available data from both the Prevaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 0.5, 95% CI 2-sided [0.41 to 0.69] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; Geometric mean fold rise = 0.7, 95% CI 2-sided [0.60 to 0.82] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 9: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; Geometric mean fold rise = 0.6, 95% CI 2-sided [0.47 to 0.76] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 5: GMFR was calculated using all participants with available data from both the Prevaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 0.8, 95% CI 2-sided [0.67 to 0.87] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; Geometric mean fold rise = 1.1, 95% CI 2-sided [0.96 to 1.30] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 12: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; Geometric mean fold rise = 0.9, 95% CI 2-sided [0.75 to 1.02] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 6A: GMFR was calculated using all participants with available data from both the Prevaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 0.6, 95% CI 2-sided [0.48 to 0.79] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 14: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; Geometric mean fold rise = 0.4, 95% CI 2-sided [0.32 to 0.46] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 15: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; Geometric mean fold rise = 1.3, 95% CI 2-sided [0.94 to 1.75] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 16: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 6B: GMFR was calculated using all participants with available data from both the Prevaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 1.7, 95% CI 2-sided [1.32 to 2.19] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 17: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; Geometric mean fold rise = 1.4, 95% CI 2-sided [1.14 to 1.60] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 18: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; Geometric mean fold rise = 1.6, 95% CI 2-sided [1.20 to 2.01] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 19: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 7F: GMFR was calculated using all participants with available data from both the Prevaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 1.7, 95% CI 2-sided [1.24 to 2.26] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 20: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 4, analysis 19]; Test type: Superiority or Other; Geometric mean fold rise = 3.1, 95% CI 2-sided [2.26 to 4.30] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 21: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 4, analysis 19]; Test type: Superiority or Other; Geometric mean fold rise = 2.0, 95% CI 2-sided [1.53 to 2.75] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 22: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 9V: GMFR was calculated using all participants with available data from both the Prevaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 2.1, 95% CI 2-sided [1.48 to 2.95] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 23: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; Geometric mean fold rise = 2.7, 95% CI 2-sided [1.97 to 3.70] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 24: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; Geometric mean fold rise = 2.9, 95% CI 2-sided [1.99 to 4.29] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 25: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 14: GMFR was calculated using all participants with available data from both the Prevaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 1.6, 95% CI 2-sided [1.23 to 2.05] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 26: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 4, analysis 25]; Test type: Superiority or Other; Geometric mean fold rise = 1.4, 95% CI 2-sided [1.18 to 1.78] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 27: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 4, analysis 25]; Test type: Superiority or Other; Geometric mean fold rise = 1.2, 95% CI 2-sided [1.04 to 1.42] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 28: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 18C: GMFR was calculated using all participants with available data from both the Prevaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 1.0, 95% CI 2-sided [0.82 to 1.19] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 29: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 4, analysis 28]; Test type: Superiority or Other; Geometric mean fold rise = 1.1, 95% CI 2-sided [0.96 to 1.29] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 30: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 4, analysis 28]; Test type: Superiority or Other; Geometric mean fold rise = 1.0, 95% CI 2-sided [0.89 to 1.20] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 31: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 19A: GMFR was calculated using all participants with available data from both the Prevaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 1.2, 95% CI 2-sided [1.07 to 1.46] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 32: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 4, analysis 31]; Test type: Superiority or Other; Geometric mean fold rise = 1.4, 95% CI 2-sided [1.24 to 1.61] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 33: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 4, analysis 31]; Test type: Superiority or Other; Geometric mean fold rise = 1.1, 95% CI 2-sided [0.96 to 1.27] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 34: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 19F: GMFR was calculated using all participants with available data from both the Prevaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rises = 2.1, 95% CI 2-sided [1.56 to 2.80] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 35: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 4, analysis 34]; Test type: Superiority or Other; Geometric mean fold rise = 2.3, 95% CI 2-sided [1.82 to 2.88] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 36: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 4, analysis 34]; Test type: Superiority or Other; Geometric mean fold rise = 1.5, 95% CI 2-sided [1.18 to 1.90] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 37: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 23F: GMFR was calculated using all participants with available data from both the Prevaccination 2 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 1.1, 95% CI 2-sided [0.89 to 1.48] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 38: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 4, analysis 37]; Test type: Superiority or Other; Geometric mean fold rise = 0.7, 95% CI 2-sided [0.63 to 0.85] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 39: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 4, analysis 37]; Test type: Superiority or Other; Geometric mean fold rise = 1.2, 95% CI 2-sided [0.99 to 1.51] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Serotype-Specific Pneumococcal OPA GMT Antibody Persistence 1 Year After Vaccination 2 Relative to Before Vaccination 2 (Parent Study 6115A1-3005; NCT00546572)
Description: as for outcome 2
Time Frame: Month 0/Year 1 (Parent Study NCT00546572), Month 1/Year 2 (Follow-up Study NCT01025336)
Population: All-Available Immunogenicity Population. N=number of participants with valid and determinate assay results for the specified serotype at both the Prevaccination 2 and 1 Year Postvaccination 2 blood draws.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior): Participants at least 70 years of age or greater previously vaccinated with 23vPS ≥5 years before enrollment in the parent study 6115A1-3005 (NCT00546572), who completed study NCT00546572 receiving 13vPnC administered as a single dose 0.5 mL IM at Year 0 (Vaccination 1) and at Year 1 (Vaccination 2)
Arm/Group | 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) | 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior)
Number analyzed (Participants) | 217 | 219
titer
  Serotype 1, Pre Vax 2 | 33 [26.4 to 41.1] | 21 [17.1 to 26.9]
  Serotype 1, 1 Year Post Vax 2 | 38 [30.7 to 47.5] | 22 [17.5 to 27.8]
  Serotype 3, Pre Vax 2 | 16 [13.2 to 19.4] | 16 [13.0 to 19.4]
  Serotype 3, 1 Year Post Vax 2 | 19 [16.2 to 23.2] | 16 [13.3 to 19.4]
  Serotype 4, Pre Vax 2 | 129 [89.0 to 186.9] | 73 [50.4 to 104.7]
  Serotype 4, 1 Year Post Vax 2 | 267 [198.8 to 358.8] | 177 [129.9 to 240.0]
  Serotype 5, Pre Vax 2 | 32 [25.0 to 41.4] | 24 [18.0 to 30.8]
  Serotype 5, 1 Year Post Vax 2 | 57 [44.5 to 73.2] | 42 [32.2 to 55.6]
  Serotype 6A, Pre Vax 2 | 279 [203.4 to 383.4] | 58 [41.9 to 81.1]
  Serotype 6A, 1 Year Post Vax 2 | 256 [191.2 to 341.9] | 113 [82.5 to 155.2]
  Serotype 6B, Pre Vax 2 | 403 [290.6 to 558.3] | 186 [131.1 to 264.3]
  Serotype 6B, 1 Year Post Vax 2 | 511 [376.9 to 693.4] | 361 [263.4 to 495.7]
  Serotype 7F, Pre Vax 2 | 66 [46.3 to 95.3] | 66 [45.5 to 95.0]
  Serotype 7F, 1 Year Post Vax 2 | 175 [127.1 to 240.3] | 111 [78.4 to 157.4]
  Serotype 9V, Pre Vax 2 | 40 [27.6 to 59.1] | 28 [19.7 to 40.6]
  Serotype 9V, 1 Year Post Vax 2 | 76 [51.6 to 112.9] | 69 [47.3 to 100.9]
  Serotype 14, Pre Vax 2 | 130 [96.1 to 176.2] | 144 [104.7 to 198.7]
  Serotype 14, 1 Year Post Vax 2 | 204 [155.6 to 268.5] | 240 [180.7 to 319.3]
  Serotype 18C, Pre Vax 2 | 436 [340.9 to 556.7] | 271 [197.8 to 371.7]
  Serotype 18C, 1 Year Post Vax 2 | 545 [438.2 to 678.0] | 360 [272.5 to 475.9]
  Serotype 19A, Pre Vax 2 | 185 [152.8 to 222.9] | 124 [97.4 to 158.3]
  Serotype 19A, 1 Year Post Vax 2 | 235 [196.4 to 282.2] | 181 [146.7 to 223.8]
  Serotype 19F, Pre Vax 2 | 121 [91.1 to 160.0] | 84 [61.6 to 115.4]
  Serotype 19F, 1 Year Post Vax 2 | 261 [204.9 to 333.7] | 159 [119.0 to 211.4]
  Serotype 23F, Pre Vax 2 | 60 [44.5 to 81.1] | 30 [22.3 to 41.0]
  Serotype 23F, 1 Year Post Vax 2 | 104 [78.0 to 137.4] | 46 [33.9 to 61.8]
Statistical Analysis 1: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Geometric mean fold rise = 1.2, 95% CI 2-sided [1.03 to 1.31] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Geometric mean fold rise = 1.0, 95% CI 2-sided [0.91 to 1.16] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; Geometric mean fold rise = 1.2, 95% CI 2-sided [1.07 to 1.37] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; Geometric mean fold rise = 1.0, 95% CI 2-sided [0.91 to 1.13] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; Geometric mean fold rise = 2.1, 95% CI 2-sided [1.60 to 2.68] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; Geometric mean fold rise = 2.4, 95% CI 2-sided [1.82 to 3.24] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; Geometric mean fold rise = 1.8, 95% CI 2-sided [1.55 to 2.03] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 8: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; Geometric mean fold rise = 1.8, 95% CI 2-sided [1.54 to 2.09] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; Geometric mean fold rise = 0.9, 95% CI 2-sided [0.79 to 1.07] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 10: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; Geometric mean fold rise = 1.9, 95% CI 2-sided [1.48 to 2.55] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; Geometric mean fold rise = 1.3, 95% CI 2-sided [1.05 to 1.53] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 12: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; Geometric mean fold rise = 1.9, 95% CI 2-sided [1.50 to 2.51] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 19]; Test type: Superiority or Other; Geometric mean fold rise = 2.6, 95% CI 2-sided [1.98 to 3.50] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 14: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 19]; Test type: Superiority or Other; Geometric mean fold rise = 1.7, 95% CI 2-sided [1.31 to 2.18] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 15: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; Geometric mean fold rise = 1.9, 95% CI 2-sided [1.37 to 2.61] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 16: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; Geometric mean fold rise = 2.4, 95% CI 2-sided [1.76 to 3.38] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 17: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 25]; Test type: Superiority or Other; Geometric mean fold rise = 1.6, 95% CI 2-sided [1.33 to 1.86] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 18: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 25]; Test type: Superiority or Other; Geometric mean fold rise = 1.7, 95% CI 2-sided [1.38 to 2.01] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 19: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 28]; Test type: Superiority or Other; Geometric mean fold rise = 1.3, 95% CI 2-sided [1.10 to 1.42] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 20: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 28]; Test type: Superiority or Other; Geometric mean fold rise = 1.3, 95% CI 2-sided [1.14 to 1.55] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 21: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 31]; Test type: Superiority or Other; Geometric mean fold rise = 1.3, 95% CI 2-sided [1.14 to 1.43] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 22: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 31]; Test type: Superiority or Other; Geometric mean fold rise = 1.5, 95% CI 2-sided [1.28 to 1.67] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 23: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 34]; Test type: Superiority or Other; Geometric mean fold rise = 2.2, 95% CI 2-sided [1.80 to 2.60] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 24: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 34]; Test type: Superiority or Other; Geometric mean fold rise = 1.9, 95% CI 2-sided [1.53 to 2.31] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 25: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 37]; Test type: Superiority or Other; Geometric mean fold rise = 1.7, 95% CI 2-sided [1.44 to 2.06] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 26: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 37]; Test type: Superiority or Other; Geometric mean fold rise = 1.5, 95% CI 2-sided [1.24 to 1.84] — [estimate comment as in outcome 3, analysis 1]

6. Secondary Outcome: Serotype-Specific Pneumococcal OPA GMT Antibody Persistence 1 Year After Vaccination 2 Relative to 1 Month After Vaccination 1 (Parent Study 6115A1-3010; NCT00574548)
Description: as for outcome 2
Time Frame: Month 1/Year 0 (Parent Study NCT00574548), Month 1/Year 2 (Follow-up Study NCT01025336)
Population: All-Available Immunogenicity Population. N=number of participants with valid and determinate assay results for the specified serotype at both the 1 Month Postvaccination 1 and 1 Year Postvaccination 2 blood draws.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC/13vPnC Group (23vPS Naïve) | 13vPnC/23vPS Group (23vPS Naïve) | 23vPS/13vPnC Group (23vPS Naïve)
Number analyzed (Participants) | 127 | 199 | 171
titer
  Serotype 1, 1 Month Post Vax 1 | 229 [176.7 to 295.9] | 228 [185.8 to 280.7] | 147 [112.6 to 192.0]
  Serotype 1, 1 Year Post Vax 2 | 54 [40.6 to 71.4] | 47 [37.5 to 60.0] | 35 [26.6 to 46.3]
  Serotype 3, 1 Month Post Vax 1 | 75 [59.1 to 95.5] | 75 [61.6 to 91.6] | 85 [69.0 to 103.9]
  Serotype 3, 1 Year Post Vax 2 | 19 [14.8 to 23.3] | 27 [22.5 to 32.8] | 18 [14.8 to 22.5]
  Serotype 4, 1 Month Post Vax 1 | 2546 [1908.6 to 3395.8] | 2575 [2075.2 to 3195.9] | 1406 [1026.6 to 1926.5]
  Serotype 4, 1 Year Post Vax 2 | 346 [242.6 to 493.7] | 405 [304.4 to 538.3] | 184 [127.1 to 267.4]
  Serotype 5, 1 Month Post Vax 1 | 153 [101.6 to 229.5] | 255 [190.1 to 341.4] | 145 [106.8 to 197.9]
  Serotype 5, 1 Year Post Vax 2 | 26 [18.5 to 37.8] | 69 [52.4 to 91.8] | 45 [33.6 to 61.0]
  Serotype 6A, 1 Month Post Vax 1 | 2757 [2027.3 to 3750.3] | 3022 [2356.7 to 3875.6] | 335 [227.3 to 494.8]
  Serotype 6A, 1 Year Post Vax 2 | 286 [195.1 to 418.1] | 235 [171.4 to 320.9] | 105 [73.1 to 152.2]
  Serotype 6B, 1 Month Post Vax 1 | 1739 [1176.0 to 2570.2] | 1969 [1512.1 to 2562.7] | 767 [545.3 to 1080.0]
  Serotype 6B, 1 Year Post Vax 2 | 855 [595.2 to 1227.5] | 697 [523.9 to 926.4] | 319 [220.5 to 462.1]
  Serotype 7F, 1 Month Post Vax 1 | 906 [590.6 to 1388.7] | 1459 [1147.2 to 1855.1] | 365 [243.8 to 546.8]
  Serotype 7F, 1 Year Post Vax 2 | 231 [148.8 to 359.6] | 398 [301.1 to 527.0] | 143 [97.9 to 208.2]
  Serotype 9V, 1 Month Post Vax 1 | 1055 [740.6 to 1502.7] | 801 [589.0 to 1090.0] | 294 [192.2 to 449.9]
  Serotype 9V, 1 Year Post Vax 2 | 203 [127.4 to 322.0] | 224 [155.1 to 322.3] | 127 [82.5 to 196.0]
  Serotype 14, 1 Month Post Vax 1 | 614 [409.0 to 921.9] | 727 [527.6 to 1000.7] | 748 [535.4 to 1045.9]
  Serotype 14, 1 Year Post Vax 2 | 387 [277.1 to 540.7] | 435 [329.4 to 575.6] | 391 [291.9 to 524.8]
  Serotype 18C, 1 Month Post Vax 1 | 1603 [1153.7 to 2226.2] | 1614 [1230.2 to 2117.7] | 888 [639.0 to 1233.2]
  Serotype 18C, 1 Year Post Vax 2 | 409 [281.0 to 596.0] | 560 [424.2 to 739.8] | 323 [227.9 to 457.0]
  Serotype 19A, 1 Month Post Vax 1 | 698 [522.4 to 932.2] | 781 [662.0 to 920.4] | 380 [296.6 to 486.6]
  Serotype 19A, 1 Year Post Vax 2 | 243 [185.7 to 319.1] | 310 [260.8 to 369.0] | 162 [126.7 to 207.7]
  Serotype 19F, 1 Month Post Vax 1 | 530 [361.7 to 775.7] | 845 [661.8 to 1079.9] | 423 [302.2 to 591.4]
  Serotype 19F, 1 Year Post Vax 2 | 239 [166.7 to 342.6] | 416 [333.0 to 519.7] | 180 [131.7 to 245.7]
  Serotype 23F, 1 Month Post Vax 1 | 339 [219.9 to 521.8] | 367 [268.3 to 501.2] | 72 [49.1 to 104.7]
  Serotype 23F, 1 Year Post Vax 2 | 105 [69.5 to 159.3] | 70 [52.0 to 95.0] | 39 [27.6 to 53.8]
Statistical Analysis 1: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 1: GMFR was calculated using all participants with available data from both the 1 Month Postvaccination 1 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.2, 95% CI 2-sided [0.19 to 0.29] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Geometric mean fold rise = 0.2, 95% CI 2-sided [0.17 to 0.25] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Geometric mean fold rise = 0.2, 95% CI 2-sided [0.20 to 0.29] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 3: GMFR was calculated using all participants with available data from both the 1 Month Postvaccination 1 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 0.2, 95% CI 2-sided [0.20 to 0.30] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; Geometric mean fold rise = 0.4, 95% CI 2-sided [0.31 to 0.42] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; Geometric mean fold rise = 0.2, 95% CI 2-sided [0.18 to 0.26] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 4: GMFR was calculated using all participants with available data from both the 1 Month Postvaccination 1 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 0.1, 95% CI 2-sided [0.10 to 0.18] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; Geometric mean fold rise = 0.2, 95% CI 2-sided [0.12 to 0.20] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; Geometric mean fold rise = 0.1, 95% CI 2-sided [0.10 to 0.18] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 5: GMFR was calculated using all participants with available data from both the 1 Month Postvaccination 1 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 0.2, 95% CI 2-sided [0.13 to 0.22] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; Geometric mean fold rise = 0.3, 95% CI 2-sided [0.22 to 0.33] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; Geometric mean fold rise = 0.3, 95% CI 2-sided [0.25 to 0.38] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 6A: GMFR was calculated using all participants with available data from both the 1 Month Postvaccination 1 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 0.1, 95% CI 2-sided [0.08 to 0.14] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 14: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; Geometric mean fold rise = 0.1, 95% CI 2-sided [0.06 to 0.10] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 15: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; Geometric mean fold rise = 0.3, 95% CI 2-sided [0.22 to 0.46] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 16: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 6B: GMFR was calculated using all participants with available data from both the 1 Month Postvaccination 1 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 0.5, 95% CI 2-sided [0.40 to 0.60] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 17: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 6, analysis 16]; Test type: Superiority or Other; Geometric mean fold rise = 0.4, 95% CI 2-sided [0.29 to 0.43] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 18: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 6, analysis 16]; Test type: Superiority or Other; Geometric mean fold rise = 0.4, 95% CI 2-sided [0.29 to 0.59] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 19: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 7F: GMFR was calculated using all participants with available data from both the 1 Month Postvaccination 1 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 0.3, 95% CI 2-sided [0.17 to 0.38] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 20: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 6, analysis 19]; Test type: Superiority or Other; Geometric mean fold rise = 0.3, 95% CI 2-sided [0.21 to 0.36] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 21: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 6, analysis 19]; Test type: Superiority or Other; Geometric mean fold rise = 0.4, 95% CI 2-sided [0.27 to 0.56] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 22: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 9V: GMFR was calculated using all participants with available data from both the 1 Month Postvaccination 1 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 0.2, 95% CI 2-sided [0.13 to 0.28] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 23: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 6, analysis 22]; Test type: Superiority or Other; Geometric mean fold rise = 0.3, 95% CI 2-sided [0.20 to 0.39] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 24: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 6, analysis 22]; Test type: Superiority or Other; Geometric mean fold rise = 0.4, 95% CI 2-sided [0.28 to 0.67] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 25: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 14: GMFR was calculated using all participants with available data from both the 1 Month Postvaccination 1 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 0.6, 95% CI 2-sided [0.48 to 0.83] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 26: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 6, analysis 25]; Test type: Superiority or Other; Geometric mean fold rise = 0.6, 95% CI 2-sided [0.49 to 0.74] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 27: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 6, analysis 25]; Test type: Superiority or Other; Geometric mean fold rise = 0.5, 95% CI 2-sided [0.42 to 0.65] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 28: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 18C: GMFR was calculated using all participants with available data from both the 1 Month Postvaccination 1 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 0.3, 95% CI 2-sided [0.20 to 0.32] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 29: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 6, analysis 28]; Test type: Superiority or Other; Geometric mean fold rise = 0.3, 95% CI 2-sided [0.28 to 0.43] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 30: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 6, analysis 28]; Test type: Superiority or Other; Geometric mean fold rise = 0.4, 95% CI 2-sided [0.29 to 0.45] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 31: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 19A: GMFR was calculated using all participants with available data from both the 1 Month Postvaccination 1 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 0.3, 95% CI 2-sided [0.30 to 0.41] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 32: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 6, analysis 31]; Test type: Superiority or Other; Geometric mean fold rise = 0.4, 95% CI 2-sided [0.35 to 0.45] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 33: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 6, analysis 31]; Test type: Superiority or Other; Geometric mean fold rise = 0.4, 95% CI 2-sided [0.36 to 0.51] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 34: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 19F: GMFR was calculated using all participants with available data from both the 1 Month Postvaccination 1 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 0.5, 95% CI 2-sided [0.35 to 0.58] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 35: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 6, analysis 34]; Test type: Superiority or Other; Geometric mean fold rise = 0.5, 95% CI 2-sided [0.39 to 0.62] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 36: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 6, analysis 34]; Test type: Superiority or Other; Geometric mean fold rise = 0.4, 95% CI 2-sided [0.34 to 0.54] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 37: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 23F: GMFR was calculated using all participants with available data from both the 1 Month Postvaccination 1 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; Geometric mean fold rise = 0.3, 95% CI 2-sided [0.23 to 0.42] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 38: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 6, analysis 37]; Test type: Superiority or Other; Geometric mean fold rise = 0.2, 95% CI 2-sided [0.15 to 0.24] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 39: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 6, analysis 37]; Test type: Superiority or Other; Geometric mean fold rise = 0.5, 95% CI 2-sided [0.42 to 0.69] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Serotype-Specific Pneumococcal OPA GMT Antibody Persistence 1 Year After Vaccination 2 Relative to 1 Month After Vaccination 1 (Parent Study 6115A1-3005; NCT00546572)
Description: as for outcome 2
Time Frame: Month 1/Year 0 (Parent Study NCT00546572), Month 1/Year 2 (Follow-up Study NCT01025336)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) | 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior)
Number analyzed (Participants) | 214 | 218
titer
  Serotype 1, 1 Month Post Vax 1 | 92 [72.4 to 118.0] | 53 [41.5 to 68.2]
  Serotype 1, 1 Year Post Vax 2 | 39 [31.5 to 48.6] | 22 [17.5 to 28.0]
  Serotype 3, 1 Month Post Vax 1 | 52 [42.2 to 63.2] | 51 [41.5 to 63.5]
  Serotype 3, 1 Year Post Vax 2 | 19 [16.2 to 23.4] | 16 [13.1 to 19.1]
  Serotype 4, 1 Month Post Vax 1 | 511 [374.5 to 697.2] | 216 [151.2 to 308.2]
  Serotype 4, 1 Year Post Vax 2 | 271 [203.9 to 361.3] | 185 [136.2 to 249.9]
  Serotype 5, 1 Month Post Vax 1 | 84 [64.7 to 108.8] | 42 [31.6 to 55.2]
  Serotype 5, 1 Year Post Vax 2 | 58 [45.6 to 75.0] | 42 [31.9 to 55.2]
  Serotype 6A, 1 Month Post Vax 1 | 975 [715.1 to 1328.4] | 106 [75.2 to 149.1]
  Serotype 6A, 1 Year Post Vax 2 | 264 [197.8 to 353.4] | 115 [84.3 to 158.2]
  Serotype 6B, 1 Month Post Vax 1 | 1331 [981.1 to 1806.1] | 465 [333.3 to 648.1]
  Serotype 6B, 1 Year Post Vax 2 | 553 [411.3 to 743.9] | 396 [289.7 to 540.2]
  Serotype 7F, 1 Month Post Vax 1 | 328 [233.5 to 459.8] | 195 [134.4 to 281.9]
  Serotype 7F, 1 Year Post Vax 2 | 165 [119.3 to 227.8] | 112 [79.2 to 159.1]
  Serotype 9V, 1 Month Post Vax 1 | 193 [131.4 to 282.8] | 102 [68.2 to 152.2]
  Serotype 9V, 1 Year Post Vax 2 | 82 [55.3 to 121.8] | 69 [46.9 to 101.2]
  Serotype 14, 1 Month Post Vax 1 | 241 [179.4 to 325.0] | 280 [203.3 to 384.3]
  Serotype 14, 1 Year Post Vax 2 | 205 [155.8 to 270.6] | 236 [175.5 to 318.0]
  Serotype 18C, 1 Month Post Vax 1 | 946 [749.2 to 1195.4] | 555 [405.8 to 759.9]
  Serotype 18C, 1 Year Post Vax 2 | 544 [435.5 to 679.5] | 370 [276.9 to 495.3]
  Serotype 19A, 1 Month Post Vax 1 | 381 [312.9 to 462.9] | 199 [157.3 to 251.4]
  Serotype 19A, 1 Year Post Vax 2 | 232 [192.7 to 279.3] | 180 [145.9 to 222.1]
  Serotype 19F, 1 Month Post Vax 1 | 407 [312.1 to 531.7] | 238 [177.4 to 320.2]
  Serotype 19F, 1 Year Post Vax 2 | 281 [219.7 to 358.5] | 158 [118.2 to 211.0]
  Serotype 23F, 1 Month Post Vax 1 | 173 [125.5 to 239.6] | 48 [35.2 to 65.6]
  Serotype 23F, 1 Year Post Vax 2 | 106 [79.7 to 141.5] | 45 [33.0 to 60.2]
Statistical Analysis 1: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Geometric mean fold rise = 0.4, 95% CI 2-sided [0.36 to 0.50] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Geometric mean fold rise = 0.4, 95% CI 2-sided [0.36 to 0.48] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; Geometric mean fold rise = 0.4, 95% CI 2-sided [0.33 to 0.44] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; Geometric mean fold rise = 0.3, 95% CI 2-sided [0.26 to 0.37] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; Geometric mean fold rise = 0.5, 95% CI 2-sided [0.42 to 0.68] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 6, analysis 7]; Test type: Superiority or Other; Geometric mean fold rise = 0.9, 95% CI 2-sided [0.64 to 1.14] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; Geometric mean fold rise = 0.7, 95% CI 2-sided [0.60 to 0.82] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; Geometric mean fold rise = 1.0, 95% CI 2-sided [0.86 to 1.18] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; Geometric mean fold rise = 0.3, 95% CI 2-sided [0.22 to 0.33] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 6, analysis 13]; Test type: Superiority or Other; Geometric mean fold rise = 1.1, 95% CI 2-sided [0.81 to 1.46] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 6, analysis 16]; Test type: Superiority or Other; Geometric mean fold rise = 0.4, 95% CI 2-sided [0.34 to 0.51] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 6, analysis 16]; Test type: Superiority or Other; Geometric mean fold rise = 0.9, 95% CI 2-sided [0.66 to 1.09] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 6, analysis 19]; Test type: Superiority or Other; Geometric mean fold rise = 0.5, 95% CI 2-sided [0.37 to 0.68] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 14: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 6, analysis 19]; Test type: Superiority or Other; Geometric mean fold rise = 0.6, 95% CI 2-sided [0.43 to 0.77] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 15: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 6, analysis 22]; Test type: Superiority or Other; Geometric mean fold rise = 0.4, 95% CI 2-sided [0.30 to 0.60] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 16: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 6, analysis 22]; Test type: Superiority or Other; Geometric mean fold rise = 0.7, 95% CI 2-sided [0.47 to 0.98] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 17: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 6, analysis 25]; Test type: Superiority or Other; Geometric mean fold rise = 0.9, 95% CI 2-sided [0.72 to 1.01] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 18: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 6, analysis 25]; Test type: Superiority or Other; Geometric mean fold rise = 0.8, 95% CI 2-sided [0.71 to 1.00] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 19: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 6, analysis 28]; Test type: Superiority or Other; Geometric mean fold rise = 0.6, 95% CI 2-sided [0.50 to 0.66] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 20: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 6, analysis 28]; Test type: Superiority or Other; Geometric mean fold rise = 0.7, 95% CI 2-sided [0.56 to 0.80] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 21: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 6, analysis 31]; Test type: Superiority or Other; Geometric mean fold rise = 0.6, 95% CI 2-sided [0.54 to 0.69] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 22: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 6, analysis 31]; Test type: Superiority or Other; Geometric mean fold rise = 0.9, 95% CI 2-sided [0.78 to 1.05] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 23: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 6, analysis 34]; Test type: Superiority or Other; Geometric mean fold rise = 0.7, 95% CI 2-sided [0.59 to 0.80] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 24: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 6, analysis 34]; Test type: Superiority or Other; Geometric mean fold rise = 0.7, 95% CI 2-sided [0.53 to 0.83] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 25: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 6, analysis 37]; Test type: Superiority or Other; Geometric mean fold rise = 0.6, 95% CI 2-sided [0.51 to 0.74] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 26: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 6, analysis 37]; Test type: Superiority or Other; Geometric mean fold rise = 0.9, 95% CI 2-sided [0.75 to 1.15] — [estimate comment as in outcome 2, analysis 1]

8. Secondary Outcome: Serotype-Specific Pneumococcal OPA GMT Antibody Persistence 1 Year After Vaccination 2 Relative to Before Vaccination 1 (Parent Study 6115A1-3010; NCT00574548)
Description: as for outcome 2
Time Frame: Month 0/Year 0 (Parent Study NCT00574548), Month 1/Year 2 (Follow-up Study NCT01025336)
Population: All-Available Immunogenicity Population. N=number of participants with valid and determinate assay results for the specified serotype at both the Prevaccination 1 and 1 Year Postvaccination 2 blood draws.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC/13vPnC Group (23vPS Naïve) | 13vPnC/23vPS Group (23vPS Naïve) | 23vPS/13vPnC Group (23vPS Naïve)
Number analyzed (Participants) | 127 | 209 | 173
titer
  Serotype 1, Pre Vax 1 | 7 [5.6 to 7.9] | 6 [5.4 to 7.1] | 7 [6.2 to 8.9]
  Serotype 1, 1 Year Post Vax 2 | 54 [40.8 to 70.4] | 52 [40.9 to 65.5] | 36 [27.0 to 46.8]
  Serotype 3, Pre Vax 1 | 6 [5.0 to 6.9] | 6 [5.3 to 7.0] | 7 [5.6 to 7.7]
  Serotype 3, 1 Year Post Vax 2 | 19 [14.9 to 23.5] | 27 [22.1 to 32.3] | 17 [14.0 to 21.3]
  Serotype 4, Pre Vax 1 | 24 [14.7 to 40.3] | 36 [23.8 to 54.0] | 31 [20.3 to 47.2]
  Serotype 4, 1 Year Post Vax 2 | 314 [208.6 to 472.1] | 323 [233.9 to 445.7] | 170 [115.4 to 249.2]
  Serotype 5, Pre Vax 1 | 5 [4.2 to 5.3] | 6 [5.2 to 6.9] | 6 [4.9 to 6.6]
  Serotype 5, 1 Year Post Vax 2 | 29 [20.4 to 41.4] | 75 [57.4 to 99.2] | 43 [31.4 to 57.6]
  Serotype 6A, Pre Vax 1 | 21 [13.5 to 31.9] | 17 [12.4 to 24.6] | 14 [10.1 to 20.4]
  Serotype 6A, 1 Year Post Vax 2 | 313 [210.4 to 464.4] | 214 [153.1 to 298.7] | 94 [64.0 to 137.6]
  Serotype 6B, Pre Vax 1 | 35 [20.6 to 58.4] | 24 [16.7 to 35.7] | 26 [17.3 to 40.1]
  Serotype 6B, 1 Year Post Vax 2 | 720 [474.8 to 1090.7] | 522 [378.0 to 719.8] | 292 [197.3 to 431.9]
  Serotype 7F, Pre Vax 1 | 7 [5.4 to 10.0] | 8 [6.3 to 10.5] | 7 [5.7 to 9.5]
  Serotype 7F, 1 Year Post Vax 2 | 238 [152.5 to 370.7] | 384 [290.3 to 508.9] | 143 [97.6 to 208.7]
  Serotype 9V, Pre Vax 1 | 15 [9.5 to 22.5] | 15 [10.7 to 21.5] | 18 [11.9 to 26.0]
  Serotype 9V, 1 Year Post Vax 2 | 187 [116.1 to 301.9] | 192 [130.6 to 283.3] | 119 [76.6 to 185.1]
  Serotype 14, Pre Vax 1 | 27 [17.6 to 42.5] | 34 [23.1 to 48.6] | 46 [30.9 to 67.1]
  Serotype 14, 1 Year Post Vax 2 | 350 [249.6 to 489.5] | 385 [286.5 to 518.5] | 366 [271.3 to 494.2]
  Serotype 18C, Pre Vax 1 | 20 [13.5 to 29.7] | 25 [17.8 to 33.8] | 33 [22.9 to 47.5]
  Serotype 18C, 1 Year Post Vax 2 | 400 [274.2 to 584.1] | 546 [415.3 to 718.0] | 324 [229.8 to 455.8]
  Serotype 19A, Pre Vax 1 | 20 [14.6 to 28.6] | 25 [19.1 to 32.9] | 21 [15.9 to 28.5]
  Serotype 19A, 1 Year Post Vax 2 | 245 [188.5 to 319.5] | 327 [273.7 to 391.0] | 162 [125.9 to 209.4]
  Serotype 19F, Pre Vax 1 | 20 [13.1 to 29.0] | 24 [17.3 to 33.4] | 16 [11.7 to 22.5]
  Serotype 19F, 1 Year Post Vax 2 | 237 [165.0 to 340.7] | 415 [332.9 to 516.2] | 186 [136.5 to 253.0]
  Serotype 23F, Pre Vax 1 | 10 [7.0 to 13.0] | 9 [7.1 to 11.2] | 7 [5.8 to 8.9]
  Serotype 23F, 1 Year Post Vax 2 | 114 [75.4 to 172.9] | 59 [43.9 to 80.6] | 34 [24.2 to 47.1]
Statistical Analysis 1: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 1: GMFR was calculated using all participants with available data from both the Prevaccination 1 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 8.0, 95% CI 2-sided [6.05 to 10.67] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; geometric mean fold rise = 8.3, 95% CI 2-sided [6.65 to 10.45] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; geometric mean fold rise = 4.8, 95% CI 2-sided [3.71 to 6.14] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 3: GMFR was calculated using all participants with available data from both the Prevaccination 1 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 3.2, 95% CI 2-sided [2.59 to 3.91] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 8, analysis 4]; Test type: Superiority or Other; geometric mean fold rise = 4.4, 95% CI 2-sided [3.67 to 5.26] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 8, analysis 4]; Test type: Superiority or Other; geometric mean fold rise = 2.6, 95% CI 2-sided [2.20 to 3.14] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 4: GMFR was calculated using all participants with available data from both the Prevaccination 1 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 12.9, 95% CI 2-sided [7.80 to 21.34] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; geometric mean fold rise = 9.0, 95% CI 2-sided [6.26 to 12.92] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; geometric mean fold rise = 5.5, 95% CI 2-sided [3.71 to 8.07] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 5: GMFR was calculated using all participants with available data from both the Prevaccination 1 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 6.2, 95% CI 2-sided [4.35 to 8.80] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 8, analysis 10]; Test type: Superiority or Other; geometric mean fold rise = 12.6, 95% CI 2-sided [9.71 to 16.30] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 8, analysis 10]; Test type: Superiority or Other; geometric mean fold rise = 7.5, 95% CI 2-sided [5.59 to 10.02] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 6A: GMFR was calculated using all participants with available data from both the Prevaccination 1 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 15.1, 95% CI 2-sided [9.56 to 23.81] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 14: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; geometric mean fold rise = 12.3, 95% CI 2-sided [8.66 to 17.38] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 15: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; geometric mean fold rise = 6.5, 95% CI 2-sided [4.29 to 9.89] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 16: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 6B: GMFR was calculated using all participants with available data from both the Prevaccination 1 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 20.8, 95% CI 2-sided [12.59 to 34.24] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 17: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 8, analysis 16]; Test type: Superiority or Other; geometric mean fold rise = 21.4, 95% CI 2-sided [14.56 to 31.46] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 18: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 8, analysis 16]; Test type: Superiority or Other; geometric mean fold rise = 11.1, 95% CI 2-sided [7.24 to 17.01] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 19: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 7F: GMFR was calculated using all participants with available data from both the Prevaccination 1 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 32.2, 95% CI 2-sided [19.75 to 52.57] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 20: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 8, analysis 19]; Test type: Superiority or Other; geometric mean fold rise = 47.2, 95% CI 2-sided [34.00 to 65.43] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 21: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 8, analysis 19]; Test type: Superiority or Other; geometric mean fold rise = 19.4, 95% CI 2-sided [12.95 to 29.17] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 22: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 9V: GMFR was calculated using all participants with available data from both the Prevaccination 1 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 12.8, 95% CI 2-sided [7.79 to 21.13] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 23: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 8, analysis 22]; Test type: Superiority or Other; geometric mean fold rise = 12.6, 95% CI 2-sided [8.56 to 18.68] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 24: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 8, analysis 22]; Test type: Superiority or Other; geometric mean fold rise = 6.8, 95% CI 2-sided [4.54 to 10.10] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 25: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 14: GMFR was calculated using all participants with available data from both the Prevaccination 1 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 12.8, 95% CI 2-sided [8.16 to 20.02] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 26: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 8, analysis 25]; Test type: Superiority or Other; geometric mean fold rise = 11.5, 95% CI 2-sided [8.15 to 16.23] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 27: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 8, analysis 25]; Test type: Superiority or Other; geometric mean fold rise = 8.0, 95% CI 2-sided [5.75 to 11.25] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 28: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 18C: GMFR was calculated using all participants with available data from both the Prevaccination 1 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 20.0, 95% CI 2-sided [12.99 to 30.76] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 29: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 8, analysis 28]; Test type: Superiority or Other; geometric mean fold rise = 22.3, 95% CI 2-sided [16.50 to 30.06] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 30: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 8, analysis 28]; Test type: Superiority or Other; geometric mean fold rise = 9.8, 95% CI 2-sided [7.07 to 13.63] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 31: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 19A: GMFR was calculated using all participants with available data from both the Prevaccination 1 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 12.0, 95% CI 2-sided [8.82 to 16.34] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 32: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 8, analysis 31]; Test type: Superiority or Other; geometric mean fold rise = 13.0, 95% CI 2-sided [10.21 to 16.66] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 33: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 8, analysis 31]; Test type: Superiority or Other; geometric mean fold rise = 7.6, 95% CI 2-sided [5.86 to 9.94] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 34: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 19F: GMFR was calculated using all participants with available data from both the Prevaccination 1 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 12.2, 95% CI 2-sided [8.05 to 18.34] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 35: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 8, analysis 34]; Test type: Superiority or Other; geometric mean fold rise = 17.2, 95% CI 2-sided [12.77 to 23.24] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 36: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 8, analysis 34]; Test type: Superiority or Other; geometric mean fold rise = 11.5, 95% CI 2-sided [8.01 to 16.45] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 37: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); Serotype 23F: GMFR was calculated using all participants with available data from both the Prevaccination 1 and 1 Year Postvaccination 2 blood draws; Test type: Superiority or Other; geometric mean fold rise = 12.0, 95% CI 2-sided [7.89 to 18.19] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 38: Comparison: 13vPnC/23vPS Group (23vPS Naïve); [analysis description as in outcome 8, analysis 37]; Test type: Superiority or Other; geometric mean fold rise = 6.7, 95% CI 2-sided [5.02 to 8.92] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 39: Comparison: 23vPS/13vPnC Group (23vPS Naïve); [analysis description as in outcome 8, analysis 37]; Test type: Superiority or Other; geometric mean fold rise = 4.7, 95% CI 2-sided [3.52 to 6.29] — [estimate comment as in outcome 2, analysis 1]

9. Secondary Outcome: Serotype-Specific Pneumococcal OPA GMT Antibody Persistence 1 Year After Vaccination 2 Relative to Before Vaccination 1 (Parent Study 6115A1-3005; NCT00546572)
Description: as for outcome 2
Time Frame: Month 0/Year 0 (Parent Study NCT00546572), Month 1/Year 2 (Follow-up Study NCT01025336)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) | 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior)
Number analyzed (Participants) | 218 | 218
titer
  Serotype 1, Pre Vax 1 | 10 [8.7 to 12.4] | 10 [7.9 to 11.5]
  Serotype 1, 1 Year Post Vax 2 | 38 [30.9 to 47.9] | 22 [17.6 to 28.1]
  Serotype 3, Pre Vax 1 | 9 [7.7 to 11.0] | 10 [8.6 to 12.2]
  Serotype 3, 1 Year Post Vax 2 | 20 [16.4 to 23.5] | 16 [12.9 to 18.7]
  Serotype 4, Pre Vax 1 | 30 [20.4 to 42.9] | 27 [19.0 to 38.7]
  Serotype 4, 1 Year Post Vax 2 | 238 [176.8 to 319.4] | 160 [117.1 to 219.2]
  Serotype 5, Pre Vax 1 | 12 [9.3 to 14.6] | 14 [10.8 to 17.6]
  Serotype 5, 1 Year Post Vax 2 | 57 [44.4 to 73.2] | 43 [32.7 to 56.7]
  Serotype 6A, Pre Vax 1 | 22 [16.0 to 29.7] | 31 [22.1 to 42.6]
  Serotype 6A, 1 Year Post Vax 2 | 259 [192.7 to 346.9] | 108 [78.4 to 148.3]
  Serotype 6B, Pre Vax 1 | 79 [54.1 to 113.9] | 123 [84.0 to 179.4]
  Serotype 6B, 1 Year Post Vax 2 | 507 [368.6 to 696.7] | 385 [278.9 to 531.9]
  Serotype 7F, Pre Vax 1 | 23 [16.4 to 32.1] | 21 [14.7 to 28.9]
  Serotype 7F, 1 Year Post Vax 2 | 169 [122.3 to 232.4] | 115 [81.7 to 163.2]
  Serotype 9V, Pre Vax 1 | 21 [14.4 to 29.9] | 23 [15.9 to 32.6]
  Serotype 9V, 1 Year Post Vax 2 | 75 [50.5 to 111.3] | 66 [45.3 to 97.4]
  Serotype 14, Pre Vax 1 | 70 [49.9 to 97.8] | 79 [55.5 to 111.2]
  Serotype 14, 1 Year Post Vax 2 | 202 [153.2 to 266.8] | 224 [167.0 to 299.6]
  Serotype 18C, Pre Vax 1 | 131 [95.8 to 178.3] | 145 [103.9 to 201.9]
  Serotype 18C, 1 Year Post Vax 2 | 530 [425.0 to 660.6] | 368 [277.8 to 488.9]
  Serotype 19A, Pre Vax 1 | 79 [62.4 to 101.1] | 66 [50.9 to 85.3]
  Serotype 19A, 1 Year Post Vax 2 | 236 [197.3 to 283.1] | 175 [141.8 to 216.8]
  Serotype 19F, Pre Vax 1 | 46 [33.2 to 62.9] | 37 [27.6 to 50.9]
  Serotype 19F, 1 Year Post Vax 2 | 272 [212.8 to 346.8] | 151 [112.6 to 201.6]
  Serotype 23F, Pre Vax 1 | 14 [11.1 to 18.4] | 16 [12.5 to 21.6]
  Serotype 23F 1 Year Post Vax 2 | 99 [74.0 to 131.6] | 45 [33.7 to 61.1]
Statistical Analysis 1: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; geometric mean fold rise = 3.7, 95% CI 2-sided [3.05 to 4.49] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; geometric mean fold rise = 2.3, 95% CI 2-sided [1.92 to 2.81] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 8, analysis 4]; Test type: Superiority or Other; geometric mean fold rise = 2.1, 95% CI 2-sided [1.83 to 2.50] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 8, analysis 4]; Test type: Superiority or Other; geometric mean fold rise = 1.5, 95% CI 2-sided [1.32 to 1.74] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; geometric mean fold rise = 8.0, 95% CI 2-sided [5.82 to 11.09] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; geometric mean fold rise = 5.9, 95% CI 2-sided [4.25 to 8.21] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 8, analysis 10]; Test type: Superiority or Other; geometric mean fold rise = 4.9, 95% CI 2-sided [3.96 to 6.00] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 8, analysis 10]; Test type: Superiority or Other; geometric mean fold rise = 3.1, 95% CI 2-sided [2.58 to 3.79] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; geometric mean fold rise = 11.9, 95% CI 2-sided [8.56 to 16.49] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; geometric mean fold rise = 3.5, 95% CI 2-sided [2.59 to 4.76] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 8, analysis 16]; Test type: Superiority or Other; geometric mean fold rise = 6.5, 95% CI 2-sided [4.61 to 9.03] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 8, analysis 16]; Test type: Superiority or Other; geometric mean fold rise = 3.1, 95% CI 2-sided [2.32 to 4.24] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 8, analysis 19]; Test type: Superiority or Other; geometric mean fold rise = 7.4, 95% CI 2-sided [5.23 to 10.33] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 14: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 8, analysis 19]; Test type: Superiority or Other; geometric mean fold rise = 5.6, 95% CI 2-sided [4.07 to 7.69] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 15: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 8, analysis 22]; Test type: Superiority or Other; geometric mean fold rise = 3.6, 95% CI 2-sided [2.50 to 5.20] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 16: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 8, analysis 22]; Test type: Superiority or Other; geometric mean fold rise = 2.9, 95% CI 2-sided [2.10 to 4.04] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 17: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 8, analysis 25]; Test type: Superiority or Other; geometric mean fold rise = 2.9, 95% CI 2-sided [2.26 to 3.71] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 18: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 8, analysis 25]; Test type: Superiority or Other; geometric mean fold rise = 2.8, 95% CI 2-sided [2.23 to 3.63] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 19: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 8, analysis 28]; Test type: Superiority or Other; geometric mean fold rise = 4.1, 95% CI 2-sided [3.16 to 5.20] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 20: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 8, analysis 28]; Test type: Superiority or Other; geometric mean fold rise = 2.5, 95% CI 2-sided [2.06 to 3.14] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 21: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 8, analysis 31]; Test type: Superiority or Other; geometric mean fold rise = 3.0, 95% CI 2-sided [2.46 to 3.60] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 22: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 8, analysis 31]; Test type: Superiority or Other; geometric mean fold rise = 2.7, 95% CI 2-sided [2.24 to 3.15] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 23: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 8, analysis 34]; Test type: Superiority or Other; geometric mean fold rise = 5.9, 95% CI 2-sided [4.55 to 7.76] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 24: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 8, analysis 34]; Test type: Superiority or Other; geometric mean fold rise = 4.0, 95% CI 2-sided [3.13 to 5.17] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 25: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 8, analysis 37]; Test type: Superiority or Other; geometric mean fold rise = 6.9, 95% CI 2-sided [5.16 to 9.25] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 26: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 8, analysis 37]; Test type: Superiority or Other; geometric mean fold rise = 2.8, 95% CI 2-sided [2.24 to 3.40] — [estimate comment as in outcome 2, analysis 1]

10. Secondary Outcome: Serotype-Specific Pneumococcal OPA GMT Antibody Persistence 1 Year After Vaccination 2 for 13vPnC/23vPS Compared to 23vPS/13vPnC (Parent Study 6115A-3010; NCT00574548)
Description: as for outcome 2
Time Frame: Month 0/Year 2 (Baseline) (Follow-up Study 6115A1-3018; NCT01025336)
Population: All-Available Immunogenicity Population. N=number of participants with a determinate OPA antibody titer to the given serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC/23vPS Group (23vPS Naïve) | 23vPS/13vPnC Group (23vPS Naïve)
Number analyzed (Participants) | 209 | 179
titer
  Serotype 1 | 52 [40.9 to 65.5] | 36 [27.1 to 46.7]
  Serotype 3 | 27 [22.2 to 32.3] | 18 [14.4 to 21.9]
  Serotype 4 | 355 [264.7 to 475.9] | 183 [127.7 to 263.2]
  Serotype 5 | 76 [58.0 to 99.7] | 44 [32.9 to 59.6]
  Serotype 6A | 225 [163.6 to 308.3] | 102 [71.4 to 146.9]
  Serotype 6B | 593 [441.4 to 797.3] | 324 [225.0 to 466.1]
  Serotype 7F | 412 [313.1 to 541.2] | 145 [100.3 to 210.7]
  Serotype 9V | 221 [154.2 to 316.0] | 129 [84.5 to 196.5]
  Serotype 14 | 416 [316.2 to 548.2] | 383 [286.9 to 510.6]
  Serotype 18C | 527 [401.7 to 690.5] | 337 [240.7 to 471.7]
  Serotype 19A | 313 [263.1 to 372.3] | 170 [134.4 to 214.8]
  Serotype 19F | 426 [343.7 to 527.7] | 195 [145.1 to 262.1]
  Serotype 23F | 64 [47.6 to 86.5] | 35 [25.6 to 48.6]
Statistical Analysis 1: Comparison: 13vPnC/23vPS Group (23vPS Naïve) vs 23vPS/13vPnC Group (23vPS Naïve); Serotype 1: Ratio of GMT (13vPnC/23vPS to 23vPS/13vPnC) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 1.5, 95% CI 2-sided [1.02 to 2.08] — CIs for the ratio are back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures [13vPnC/23vPS-23vPS/13vPnC)]
Statistical Analysis 2: Comparison: 13vPnC/23vPS Group (23vPS Naïve) vs 23vPS/13vPnC Group (23vPS Naïve); Serotype 3: Ratio of GMT (13vPnC/23vPS to 23vPS/13vPnC) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio = 1.5, 95% CI 2-sided [1.14 to 1.99] — CIs for the ratio are back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures [(13vPnC/23vPS-23vPS/13vPnC)]
Statistical Analysis 3: Comparison: 13vPnC/23vPS Group (23vPS Naïve) vs 23vPS/13vPnC Group (23vPS Naïve); Serotype 4: Ratio of GMT (13vPnC/23vPS to 23vPS/13vPnC) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio = 1.9, 95% CI 2-sided [1.22 to 3.06] — [estimate comment as in outcome 10, analysis 2]
Statistical Analysis 4: Comparison: 23vPS/13vPnC Group (23vPS Naïve); Serotype 5: Ratio of GMT (13vPnC/23vPS to 23vPS/13vPnC) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio = 1.7, 95% CI 2-sided [1.15 to 2.56] — [estimate comment as in outcome 10, analysis 2]
Statistical Analysis 5: Comparison: 13vPnC/23vPS Group (23vPS Naïve) vs 23vPS/13vPnC Group (23vPS Naïve); Serotype 6A: Ratio of GMT (13vPnC/23vPS to 23vPS/13vPnC) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio = 2.2, 95% CI 2-sided [1.36 to 3.53] — [estimate comment as in outcome 10, analysis 2]
Statistical Analysis 6: Comparison: 13vPnC/23vPS Group (23vPS Naïve) vs 23vPS/13vPnC Group (23vPS Naïve); Serotype 6B: Ratio of GMT (13vPnC/23vPS to 23vPS/13vPnC) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio = 1.8, 95% CI 2-sided [1.15 to 2.91] — [estimate comment as in outcome 10, analysis 2]
Statistical Analysis 7: Comparison: 13vPnC/23vPS Group (23vPS Naïve); Serotype 7F: Ratio of GMT (13vPnC/23vPS to 23vPS/13vPnC) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio = 2.8, 95% CI 2-sided [1.80 to 4.44] — [estimate comment as in outcome 10, analysis 2]
Statistical Analysis 8: Comparison: 13vPnC/23vPS Group (23vPS Naïve) vs 23vPS/13vPnC Group (23vPS Naïve); Serotype 9V: Ratio of GMT (13vPnC/23vPS to 23vPS/13vPnC) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio = 1.7, 95% CI 2-sided [0.99 to 2.96] — [estimate comment as in outcome 10, analysis 2]
Statistical Analysis 9: Comparison: 13vPnC/23vPS Group (23vPS Naïve) vs 23vPS/13vPnC Group (23vPS Naïve); Serotype 14: Ratio of GMT (13vPnC/23vPS to 23vPS/13vPnC) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio = 1.1, 95% CI 2-sided [0.73 to 1.62] — [estimate comment as in outcome 10, analysis 2]
Statistical Analysis 10: Comparison: 13vPnC/23vPS Group (23vPS Naïve) vs 23vPS/13vPnC Group (23vPS Naïve); Serotype 18C: Ratio of GMT (13vPnC/23vPS to 23vPS/13vPnC) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio = 1.6, 95% CI 2-sided [1.02 to 2.39] — [estimate comment as in outcome 10, analysis 2]
Statistical Analysis 11: Comparison: 13vPnC/23vPS Group (23vPS Naïve) vs 23vPS/13vPnC Group (23vPS Naïve); Serotype 19A: Ratio of GMT (13vPnC/23vPS to 23vPS/13vPnC) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio = 1.8, 95% CI 2-sided [1.38 to 2.45] — [estimate comment as in outcome 10, analysis 2]
Statistical Analysis 12: Comparison: 13vPnC/23vPS Group (23vPS Naïve) vs 23vPS/13vPnC Group (23vPS Naïve); Serotype 19F: Ratio of GMT (13vPnC/23vPS to 23vPS/13vPnC) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio = 2.2, 95% CI 2-sided [1.53 to 3.12] — [estimate comment as in outcome 10, analysis 2]
Statistical Analysis 13: Comparison: 13vPnC/23vPS Group (23vPS Naïve) vs 23vPS/13vPnC Group (23vPS Naïve); Serotype 23F: Ratio of GMT (13vPnC/23vPS to 23vPS/13vPnC) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio = 1.8, 95% CI 2-sided [1.18 to 2.82] — [estimate comment as in outcome 10, analysis 2]

11. Secondary Outcome: Serotype-Specific Pneumococcal OPA GMT Antibody Persistence 1 Year After Vaccination 2 for 13vPnC/13vPnC Compared to 23vPS/13vPnC (Parent Study 6115A1-3010; NCT00574548)
Description: as for outcome 2
Time Frame: Month 0/Year 2 (Baseline) (Follow-up Study 6115A1-3018; NCT01025336)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC/13vPnC Group (23vPS Naïve) | 23vPS/13vPnC Group (23vPS Naïve)
Number analyzed (Participants) | 129 | 179
titer
  Serotype 1 | 54 [40.8 to 71.0] | 36 [27.1 to 46.7]
  Serotype 3 | 19 [15.0 to 23.5] | 18 [14.4 to 21.9]
  Serotype 4 | 328 [229.0 to 469.0] | 183 [127.7 to 263.2]
  Serotype 5 | 29 [20.4 to 41.4] | 44 [32.9 to 59.6]
  Serotype 6A | 316 [216.5 to 461.2] | 102 [71.4 to 146.9]
  Serotype 6B | 785 [540.6 to 1140.2] | 324 [225.0 to 466.1]
  Serotype 7F | 247 [160.4 to 380.9] | 145 [100.3 to 210.7]
  Serotype 9V | 211 [134.3 to 330.9] | 129 [84.5 to 196.5]
  Serotype 14 | 379 [273.6 to 526.2] | 383 [286.9 to 510.6]
  Serotype 18C | 393 [271.3 to 569.3] | 337 [240.7 to 471.7]
  Serotype 19A | 244 [189.1 to 314.1] | 170 [134.4 to 214.8]
  Serotype 19F | 256 [182.4 to 359.0] | 195 [145.1 to 262.1]
  Serotype 23F | 110 [73.9 to 165.0] | 35 [25.6 to 48.6]
Statistical Analysis 1: Comparison: 13vPnC/13vPnC Group (23vPS Naïve) vs 23vPS/13vPnC Group (23vPS Naïve); Serotype 1: Ratio of GMT (13vPnC/13vPnC to 23vPS/13vPnC) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 1.5, 95% CI 2-sided [1.02 to 2.25] — CIs for the ratio are back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures [(13vPnC/13vPnC - 23vPS/13vPnC)]
Statistical Analysis 2: Comparison: 13vPnC/13vPnC Group (23vPS Naïve) vs 23vPS/13vPnC Group (23vPS Naïve); Serotype 3: Ratio of GMT (13vPnC/13vPnC to 23vPS/13vPnC) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 1.1, 95% CI 2-sided [0.78 to 1.44] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC/13vPnC Group (23vPS Naïve) vs 23vPS/13vPnC Group (23vPS Naïve); Serotype 4: Ratio of GMT (13vPnC/13vPnC to 23vPS/13vPnC) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 1.8, 95% CI 2-sided [1.06 to 3.00] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC/13vPnC Group (23vPS Naïve) vs 23vPS/13vPnC Group (23vPS Naïve); Serotype 5: Ratio of GMT (13vPnC/13vPnC to 23vPS/13vPnC) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 0.7, 95% CI 2-sided [0.41 to 1.04] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC/13vPnC Group (23vPS Naïve) vs 23vPS/13vPnC Group (23vPS Naïve); Serotype 6A: Ratio of GMT (13vPnC/13vPnC to 23vPS/13vPnC) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 3.1, 95% CI 2-sided [1.82 to 5.24] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: 13vPnC/13vPnC Group (23vPS Naïve) vs 23vPS/13vPnC Group (23vPS Naïve); Serotype 6B: Ratio of GMT (13vPnC/13vPnC to 23vPS/13vPnC) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 2.4, 95% CI 2-sided [1.43 to 4.11] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC/13vPnC Group (23vPS Naïve) vs 23vPS/13vPnC Group (23vPS Naïve); Serotype 7F: Ratio of GMT (13vPnC/13vPnC to 23vPS/13vPnC) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 1.7, 95% CI 2-sided [0.96 to 3.00] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC/13vPnC Group (23vPS Naïve) vs 23vPS/13vPnC Group (23vPS Naïve); Serotype 9V: Ratio of GMT (13vPnC/13vPnC to 23vPS/13vPnC) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 1.6, 95% CI 2-sided [0.88 to 3.04] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC/13vPnC Group (23vPS Naïve) vs 23vPS/13vPnC Group (23vPS Naïve); Serotype 14: Ratio of GMT (13vPnC/13vPnC to 23vPS/13vPnC) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 1.0, 95% CI 2-sided [0.64 to 1.54] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC/13vPnC Group (23vPS Naïve) vs 23vPS/13vPnC Group (23vPS Naïve); Serotype 18C: Ratio of GMT (13vPnC/13vPnC to 23vPS/13vPnC) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 1.2, 95% CI 2-sided [0.71 to 1.93] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC/13vPnC Group (23vPS Naïve) vs 23vPS/13vPnC Group (23vPS Naïve); Serotype 19A: Ratio of GMT (13vPnC/13vPnC to 23vPS/13vPnC) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 1.4, 95% CI 2-sided [1.01 to 2.04] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 12: Comparison: 13vPnC/13vPnC Group (23vPS Naïve) vs 23vPS/13vPnC Group (23vPS Naïve); Serotype 19F: Ratio of GMT (13vPnC/13vPnC to 23vPS/13vPnC) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 1.3, 95% CI 2-sided [0.84 to 2.06] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC/13vPnC Group (23vPS Naïve) vs 23vPS/13vPnC Group (23vPS Naïve); Serotype 23F: Ratio of GMT (13vPnC/13vPnC to 23vPS/13vPnC) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 3.1, 95% CI 2-sided [1.89 to 5.20] — [estimate comment as in outcome 11, analysis 1]

12. Secondary Outcome: Serotype-Specific Pneumococcal OPA GMT Antibody Persistence 1 Year After Vaccination 2 for 13vPnC/13vPnC Compared to 13vPnC/23vPS (Parent Study 6115A1-3010; NCT00574548)
Description: as for outcome 2
Time Frame: Month 0/Year 2 (Baseline) (Follow-up Study 6115A1-3018; NCT01025336)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC/13vPnC Group (23vPS Naïve) | 13vPnC/23vPS Group (23vPS Naïve)
Number analyzed (Participants) | 129 | 209
titer
  Serotype 1 | 54 [40.8 to 71.0] | 52 [40.9 to 65.5]
  Serotype 3 | 19 [15.0 to 23.5] | 27 [22.2 to 32.3]
  Serotype 4 | 328 [229.0 to 469.0] | 355 [264.7 to 475.9]
  Serotype 5 | 29 [20.4 to 41.4] | 76 [58.0 to 99.7]
  Serotype 6A | 316 [216.5 to 461.2] | 225 [163.6 to 308.3]
  Serotype 6B | 785 [540.6 to 1140.2] | 593 [441.4 to 797.3]
  Serotype 7F | 247 [160.4 to 380.9] | 412 [313.1 to 541.2]
  Serotype 9V | 211 [134.3 to 330.9] | 221 [154.2 to 316.0]
  Serotype 14 | 379 [273.6 to 526.2] | 416 [316.2 to 548.2]
  Serotype 18C | 393 [271.3 to 569.3] | 527 [401.7 to 690.5]
  Serotype 19A | 244 [189.1 to 314.1] | 313 [263.1 to 372.3]
  Serotype 19F | 256 [182.4 to 359.0] | 426 [343.7 to 527.7]
  Serotype 23F | 110 [73.9 to 165.0] | 64 [47.6 to 86.5]
Statistical Analysis 1: Comparison: 13vPnC/13vPnC Group (23vPS Naïve) vs 13vPnC/23vPS Group (23vPS Naïve); Serotype 1: Ratio of GMT (13vPnC/13vPnC to 13vPnC/23vPS) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 1.0, 95% CI 2-sided [0.72 to 1.51] — CIs for the ratio are back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures [(13vPnC/13vPnC - 13vPnC/23vPS)]
Statistical Analysis 2: Comparison: 13vPnC/13vPnC Group (23vPS Naïve) vs 13vPnC/23vPS Group (23vPS Naïve); Serotype 3: Ratio of GMT (13vPnC/13vPnC to 13vPnC/23vPS) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 0.7, 95% CI 2-sided [0.52 to 0.94] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC/13vPnC Group (23vPS Naïve) vs 13vPnC/23vPS Group (23vPS Naïve); Serotype 4: Ratio of GMT (13vPnC/13vPnC to 13vPnC/23vPS) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 0.9, 95% CI 2-sided [0.58 to 1.47] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC/13vPnC Group (23vPS Naïve) vs 13vPnC/23vPS Group (23vPS Naïve); Serotype 5: Ratio of GMT (13vPnC/13vPnC to 13vPnC/23vPS) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 0.4, 95% CI 2-sided [0.25 to 0.59] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC/13vPnC Group (23vPS Naïve) vs 13vPnC/23vPS Group (23vPS Naïve); Serotype 6A: Ratio of GMT (13vPnC/13vPnC to 13vPnC/23vPS) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 1.4, 95% CI 2-sided [0.85 to 2.32] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 6: Comparison: 13vPnC/13vPnC Group (23vPS Naïve) vs 13vPnC/23vPS Group (23vPS Naïve); Serotype 6B: Ratio of GMT (13vPnC/13vPnC to 13vPnC/23vPS) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 1.3, 95% CI 2-sided [0.82 to 2.13] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC/13vPnC Group (23vPS Naïve) vs 13vPnC/23vPS Group (23vPS Naïve); Serotype 7F: Ratio of GMT (13vPnC/13vPnC to 13vPnC/23vPS) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 0.6, 95% CI 2-sided [0.37 to 0.97] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC/13vPnC Group (23vPS Naïve) vs 13vPnC/23vPS Group (23vPS Naïve); Serotype 9V: Ratio of GMT (13vPnC/13vPnC to 13vPnC/23vPS) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 1.0, 95% CI 2-sided [0.54 to 1.70] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC/13vPnC Group (23vPS Naïve) vs 13vPnC/23vPS Group (23vPS Naïve); Serotype 14: Ratio of GMT (13vPnC/13vPnC to 13vPnC/23vPS) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 0.9, 95% CI 2-sided [0.59 to 1.41] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC/13vPnC Group (23vPS Naïve) vs 13vPnC/23vPS Group (23vPS Naïve); Serotype 18C: Ratio of GMT (13vPnC/13vPnC to 13vPnC/23vPS) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 0.7, 95% CI 2-sided [0.48 to 1.17] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC/13vPnC Group (23vPS Naïve) vs 13vPnC/23vPS Group (23vPS Naïve); Serotype 19A: Ratio of GMT (13vPnC/13vPnC to 13vPnC/23vPS) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 0.8, 95% CI 2-sided [0.58 to 1.05] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 12: Comparison: 13vPnC/13vPnC Group (23vPS Naïve) vs 13vPnC/23vPS Group (23vPS Naïve); Serotype 19F: Ratio of GMT (13vPnC/13vPnC to 13vPnC/23vPS) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 0.6, 95% CI 2-sided [0.41 to 0.88] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC/13vPnC Group (23vPS Naïve) vs 13vPnC/23vPS Group (23vPS Naïve); Serotype 23F: Ratio of GMT (13vPnC/13vPnC to 13vPnC/23vPS) was calculated by back transforming the mean difference between vaccine sequence on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 1.7, 95% CI 2-sided [1.05 to 2.81] — [estimate comment as in outcome 12, analysis 1]

13. Secondary Outcome: Serotype-Specific Pneumococcal OPA GMT Antibody Persistence 1 Year After Vaccination 2 for 13vPnC/13vPnC Compared to 23vPS/13vPnC (Parent Study 6115A1-3005; NCT00546572)
Description: as for outcome 2
Time Frame: Month 0/Year 2 (Baseline) (Follow-up Study 6115A1-3018; NCT01025336)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) | 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior)
Number analyzed (Participants) | 220 | 222
titer
  Serotype 1 | 38 [30.9 to 47.9] | 22 [17.5 to 27.8]
  Serotype 3 | 20 [16.5 to 23.4] | 16 [13.3 to 19.2]
  Serotype 4 | 265 [200.8 to 348.5] | 172 [129.0 to 230.1]
  Serotype 5 | 58 [45.1 to 74.1] | 42 [32.2 to 55.6]
  Serotype 6A | 250 [187.3 to 334.0] | 115 [84.5 to 156.8]
  Serotype 6B | 510 [378.2 to 686.4] | 381 [281.9 to 513.9]
  Serotype 7F | 173 [126.0 to 237.5] | 115 [81.6 to 160.9]
  Serotype 9V | 81 [55.1 to 117.9] | 68 [47.4 to 98.5]
  Serotype 14 | 202 [154.6 to 265.0] | 240 [181.0 to 317.0]
  Serotype 18C | 540 [435.5 to 668.5] | 360 [273.6 to 474.5]
  Serotype 19A | 232 [193.2 to 278.1] | 181 [146.7 to 222.9]
  Serotype 19F | 277 [218.6 to 351.7] | 158 [119.3 to 209.9]
  Serotype 23F | 103 [78.0 to 135.0] | 45 [33.5 to 69.6]
Statistical Analysis 1: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Ratio of GMT = 1.7, 95% CI 2-sided [1.27 to 2.40] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 11, analysis 2]; Test type: Superiority or Other; Ratio of GMT = 1.2, 95% CI 2-sided [0.95 to 1.59] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 11, analysis 3]; Test type: Superiority or Other; Ratio of GMT = 1.5, 95% CI 2-sided [1.03 to 2.29] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 11, analysis 4]; Test type: Superiority or Other; Ratio of GMT = 1.4, 95% CI 2-sided [0.95 to 1.97] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 11, analysis 5]; Test type: Superiority or Other; Ratio of GMT = 2.2, 95% CI 2-sided [1.42 to 3.31] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 11, analysis 6]; Test type: Superiority or Other; Ratio of GMT = 1.3, 95% CI 2-sided [0.88 to 2.04] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 11, analysis 7]; Test type: Superiority or Other; Ratio of GMT = 1.5, 95% CI 2-sided [0.95 to 2.40] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 11, analysis 8]; Test type: Superiority or Other; Ratio of GMT = 1.2, 95% CI 2-sided [0.70 to 1.99] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 11, analysis 9]; Test type: Superiority or Other; Ratio of GMT = 0.8, 95% CI 2-sided [0.57 to 1.25] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 11, analysis 10]; Test type: Superiority or Other; Ratio of GMT = 1.5, 95% CI 2-sided [1.06 to 2.12] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 11, analysis 11]; Test type: Superiority or Other; Ratio of GMT = 1.3, 95% CI 2-sided [0.97 to 1.69] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 12: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 11, analysis 12]; Test type: Superiority or Other; Ratio of GMT = 1.8, 95% CI 2-sided [1.21 to 2.53] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 11, analysis 13]; Test type: Superiority or Other; Ratio of GMT = 2.3, 95% CI 2-sided [1.54 to 3.42] — [estimate comment as in outcome 11, analysis 1]

14. Secondary Outcome: Serotype-Specific Pneumococcal OPA GMT Antibody Persistence for 13vPnC/23vPS 1 Year After Vaccination 2 Compared to 23vPS 1 Year After Vaccination 1 (Parent Study 6115A1-3010; NCT00574548)
Description: as for outcome 2
Time Frame: Month 0/Year 1 (Parent Study NCT00574548), Month 0/Year 2 (Baseline) (Follow-up Study 6115A1-3018; NCT01025336)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- 23vPS (23vPS Naïve): Participants aged 60 to 64 years old who had never been vaccinated with 23vPS prior to enrollment into the parent study 6115A1-3010 (NCT00574548), who completed study NCT00574548 receiving 23vPS administered as a single dose 0.5 mL IM at Year 0 (Vaccination 1) and 13vPnC administered as a single dose 0.5 mL IM at Year 1 (Vaccination 2).
Arm/Group | 13vPnC/23vPS Group (23vPS Naïve) | 23vPS (23vPS Naïve)
Number analyzed (Participants) | 209 | 175
titer
  Serotype 1 | 52 [40.9 to 65.5] | 45 [34.5 to 59.8]
  Serotype 3 | 27 [22.2 to 32.3] | 26 [20.4 to 32.5]
  Serotype 4 | 355 [264.7 to 475.9] | 332 [231.8 to 476.2]
  Serotype 5 | 76 [58.0 to 99.7] | 49 [36.4 to 66.9]
  Serotype 6A | 225 [163.6 to 308.3] | 82 [54.6 to 122.4]
  Serotype 6B | 593 [441.4 to 797.3] | 162 [108.9 to 241.6]
  Serotype 7F | 412 [313.1 to 541.2] | 66 [44.1 to 100.1]
  Serotype 9V | 221 [154.2 to 316.0] | 52 [33.7 to 80.3]
  Serotype 14 | 416 [316.2 to 548.2] | 302 [214.2 to 425.3]
  Serotype 18C | 527 [401.7 to 690.5] | 319 [222.5 to 457.3]
  Serotype 19A | 313 [263.1 to 372.3] | 153 [117.3 to 199.5]
  Serotype 19F | 426 [343.7 to 527.7] | 125 [88.8 to 176.5]
  Serotype 23F | 64 [47.6 to 86.5] | 30 [21.2 to 42.1]
Statistical Analysis 1: Comparison: 13vPnC/23vPS Group (23vPS Naïve) vs 23vPS (23vPS Naïve); Serotype 1: Ratio of GMT (13vPnC/23vPS to 23vPS) was calculated by back transforming the mean difference between vaccine sequence/group on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 1.1, 95% CI 2-sided [0.80 to 1.63] — CIs for the ratio are back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures [(13vPnC/23vPS - 23vPS)]
Statistical Analysis 2: Comparison: 13vPnC/23vPS Group (23vPS Naïve) vs 23vPS (23vPS Naïve); Serotype 3: Ratio of GMT (13vPnC/23vPS to 23vPS) was calculated by back transforming the mean difference between vaccine sequence/group on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 1.0, 95% CI 2-sided [0.77 to 1.39] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC/23vPS Group (23vPS Naïve) vs 23vPS (23vPS Naïve); Serotype 4: Ratio of GMT (13vPnC/23vPS to 23vPS) was calculated by back transforming the mean difference between vaccine sequence/group on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 1.1, 95% CI 2-sided [0.68 to 1.69] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC/23vPS Group (23vPS Naïve) vs 23vPS (23vPS Naïve); Serotype 5: Ratio of GMT (13vPnC/23vPS to 23vPS) was calculated by back transforming the mean difference between vaccine sequence/group on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 1.5, 95% CI 2-sided [1.03 to 2.31] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC/23vPS Group (23vPS Naïve) vs 23vPS (23vPS Naïve); Serotype 6A: Ratio of GMT (13vPnC/23vPS to 23vPS) was calculated by back transforming the mean difference between vaccine sequence/group on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 2.7, 95% CI 2-sided [1.66 to 4.55] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 6: Comparison: 13vPnC/23vPS Group (23vPS Naïve) vs 23vPS (23vPS Naïve); Serotype 6B: Ratio of GMT (13vPnC/23vPS to 23vPS) was calculated by back transforming the mean difference between vaccine sequence/group on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 3.7, 95% CI 2-sided [2.25 to 5.94] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC/23vPS Group (23vPS Naïve) vs 23vPS (23vPS Naïve); Serotype 7F: Ratio of GMT (13vPnC/23vPS to 23vPS) was calculated by back transforming the mean difference between vaccine sequence/group on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 6.2, 95% CI 2-sided [3.85 to 9.98] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC/23vPS Group (23vPS Naïve) vs 23vPS (23vPS Naïve); Serotype 9V: Ratio of GMT (13vPnC/23vPS to 23vPS) was calculated by back transforming the mean difference between vaccine sequence/group on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 4.2, 95% CI 2-sided [2.43 to 7.40] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC/23vPS Group (23vPS Naïve) vs 23vPS (23vPS Naïve); Serotype 14: Ratio of GMT (13vPnC/23vPS to 23vPS) was calculated by back transforming the mean difference between vaccine sequence/group on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 1.4, 95% CI 2-sided [0.89 to 2.13] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC/23vPS Group (23vPS Naïve) vs 23vPS (23vPS Naïve); Serotype 18C: Ratio of GMT (13vPnC/23vPS to 23vPS) was calculated by back transforming the mean difference between vaccine sequence/group on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 1.7, 95% CI 2-sided [1.06 to 2.57] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC/23vPS Group (23vPS Naïve) vs 23vPS (23vPS Naïve); Serotype 19A: Ratio of GMT (13vPnC/23vPS to 23vPS) was calculated by back transforming the mean difference between vaccine sequence/group on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 2.0, 95% CI 2-sided [1.50 to 2.78] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 12: Comparison: 13vPnC/23vPS Group (23vPS Naïve) vs 23vPS (23vPS Naïve); Serotype 19F: Ratio of GMT (13vPnC/23vPS to 23vPS) was calculated by back transforming the mean difference between vaccine sequence/group on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 3.4, 95% CI 2-sided [2.30 to 5.04] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC/23vPS Group (23vPS Naïve) vs 23vPS (23vPS Naïve); Serotype 23F: Ratio of GMT (13vPnC/23vPS to 23vPS) was calculated by back transforming the mean difference between vaccine sequence/group on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 2.1, 95% CI 2-sided [1.37 to 3.37] — [estimate comment as in outcome 14, analysis 1]

15. Secondary Outcome: Serotype-Specific Pneumococcal OPA GMT Antibody Persistence for 23vPS/13vPnC 1 Year After Vaccination 2 Compared to 13vPnC 1 Year After Vaccination 1 (Parent Study 6115A1-3010; NCT00574548)
Description: as for outcome 2
Time Frame: Month 0/Year 1 (Parent Study NCT00574548), Month 0/Year 2 (Baseline) (Follow-up Study 6115A1-3018; NCT01025336)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- 13vPnC (23vPS Naïve): Participants aged 60 to 64 years old who had never received 23vPS prior to enrollment into the parent study 6115A1-3010 (NCT00574548), completed study NCT00574548 receiving 13vPnC administered as a single dose 0.5 mL IM at Year 0 (Vaccination 1) and either 13vPnC or 23vPS administered as a single dose 0.5 mL IM at Year 1 (Vaccination 2) (both 13vPnC/13vPnC and 13vPnC/23vPS dose groups)
Arm/Group | 23vPS/13vPnC Group (23vPS Naïve) | 13vPnC (23vPS Naïve)
Number analyzed (Participants) | 179 | 332
titer
  Serotype 1 | 36 [27.1 to 46.7] | 54 [45.4 to 65.0]
  Serotype 3 | 18 [14.4 to 21.9] | 21 [18.1 to 24.9]
  Serotype 4 | 183 [127.7 to 263.2] | 622 [496.9 to 777.7]
  Serotype 5 | 44 [32.9 to 59.6] | 52 [40.9 to 64.8]
  Serotype 6A | 102 [71.4 to 146.9] | 597 [466.8 to 764.7]
  Serotype 6B | 324 [225.0 to 466.1] | 420 [320.2 to 552.0]
  Serotype 7F | 145 [100.3 to 210.7] | 133 [99.6 to 177.8]
  Serotype 9V | 129 [84.5 to 196.5] | 85 [62.7 to 115.4]
  Serotype 14 | 383 [286.9 to 510.6] | 250 [193.5 to 324.2]
  Serotype 18C | 337 [240.7 to 471.7] | 439 [349.8 to 551.0]
  Serotype 19A | 170 [134.4 to 214.8] | 208 [175.9 to 245.7]
  Serotype 19F | 195 [145.1 to 262.1] | 147 [115.1 to 187.7]
  Serotype 23F | 35 [25.6 to 48.6] | 90 [69.9 to 116.6]
Statistical Analysis 1: Comparison: 23vPS/13vPnC Group (23vPS Naïve) vs 13vPnC (23vPS Naïve); Serotype 1: Ratio of GMT (23vPs/13vPnC to 13vPnC) was calculated by back transforming the mean difference between vaccine sequence/group on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 0.7, 95% CI 2-sided [0.48 to 0.90] — CIs for the ratio are back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures [(23vPS/13vPnC - 13vPnC)]
Statistical Analysis 2: Comparison: 23vPS/13vPnC Group (23vPS Naïve) vs 13vPnC (23vPS Naïve); Serotype 3: Ratio of GMT (23vPs/13vPnC to 13vPnC) was calculated by back transforming the mean difference between vaccine sequence/group on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 0.8, 95% CI 2-sided [0.64 to 1.09] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 3: Comparison: 23vPS/13vPnC Group (23vPS Naïve) vs 13vPnC (23vPS Naïve); Serotype 4: Ratio of GMT (23vPs/13vPnC to 13vPnC) was calculated by back transforming the mean difference between vaccine sequence/group on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 0.3, 95% CI 2-sided [0.20 to 0.44] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 4: Comparison: 23vPS/13vPnC Group (23vPS Naïve) vs 13vPnC (23vPS Naïve); Serotype 5: Ratio of GMT (23vPs/13vPnC to 13vPnC) was calculated by back transforming the mean difference between vaccine sequence/group on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 0.9, 95% CI 2-sided [0.59 to 1.26] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 5: Comparison: 23vPS/13vPnC Group (23vPS Naïve) vs 13vPnC (23vPS Naïve); Serotype 6A: Ratio of GMT (23vPs/13vPnC to 13vPnC) was calculated by back transforming the mean difference between vaccine sequence/group on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 0.2, 95% CI 2-sided [0.11 to 0.26] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 6: Comparison: 23vPS/13vPnC Group (23vPS Naïve) vs 13vPnC (23vPS Naïve); Serotype 6B: Ratio of GMT (23vPs/13vPnC to 13vPnC) was calculated by back transforming the mean difference between vaccine sequence/group on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 0.8, 95% CI 2-sided [0.49 to 1.22] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 7: Comparison: 23vPS/13vPnC Group (23vPS Naïve) vs 13vPnC (23vPS Naïve); Serotype 7F: Ratio of GMT (23vPs/13vPnC to 13vPnC) was calculated by back transforming the mean difference between vaccine sequence/group on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 1.1, 95% CI 2-sided [0.68 to 1.76] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 8: Comparison: 23vPS/13vPnC Group (23vPS Naïve) vs 13vPnC (23vPS Naïve); Serotype 9V: Ratio of GMT (23vPs/13vPnC to 13vPnC) was calculated by back transforming the mean difference between vaccine sequence/group on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 1.5, 95% CI 2-sided [0.90 to 2.55] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 9: Comparison: 23vPS/13vPnC Group (23vPS Naïve) vs 13vPnC (23vPS Naïve); Serotype 14: Ratio of GMT (23vPs/13vPnC to 13vPnC) was calculated by back transforming the mean difference between vaccine sequence/group on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 1.5, 95% CI 2-sided [1.02 to 2.30] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 10: Comparison: 23vPS/13vPnC Group (23vPS Naïve) vs 13vPnC (23vPS Naïve); Serotype 18C: Ratio of GMT (23vPs/13vPnC to 13vPnC) was calculated by back transforming the mean difference between vaccine sequence/group on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 0.8, 95% CI 2-sided [0.52 to 1.14] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 11: Comparison: 23vPS/13vPnC Group (23vPS Naïve) vs 13vPnC (23vPS Naïve); Serotype 19A: Ratio of GMT (23vPs/13vPnC to 13vPnC) was calculated by back transforming the mean difference between vaccine sequence/group on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 0.8, 95% CI 2-sided [0.62 to 1.08] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 12: Comparison: 23vPS/13vPnC Group (23vPS Naïve) vs 13vPnC (23vPS Naïve); Serotype 19F: Ratio of GMT (23vPs/13vPnC to 13vPnC) was calculated by back transforming the mean difference between vaccine sequence/group on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 1.3, 95% CI 2-sided [0.89 to 1.98] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 13: Comparison: 23vPS/13vPnC Group (23vPS Naïve) vs 13vPnC (23vPS Naïve); Serotype 23F: Ratio of GMT (23vPs/13vPnC to 13vPnC) was calculated by back transforming the mean difference between vaccine sequence/group on the logarithmic scale; Test type: Superiority or Other; Ratio of GMT = 0.4, 95% CI 2-sided [0.26 to 0.59] — [estimate comment as in outcome 15, analysis 1]

16. Secondary Outcome: Serotype-Specific Pneumococcal OPA GMT Antibody Persistence for 13vPnC/13vPnC 1 Year After Vaccination 2 Compared to 13vPnC/13vPnC Before Vaccination 2 (Parent Study 6115A1-3010; NCT00574548)
Description: as for outcome 2
Time Frame: Month 0/Year 1 (Parent Study NCT00574548), Month 0/Year 2 (Baseline) (Follow-up Study 6115A1-3018; NCT01025336)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC/13vPnC Group (23vPS Naïve)
Number analyzed (Participants) | 124
titer
  Serotype 1, Pre Vax 2 | 52 [38.2 to 69.5]
  Serotype 1, 1 Year Post Vax 2 | 52 [39.6 to 69.0]
  Serotype 3, Pre Vax 2 | 19 [14.5 to 24.1]
  Serotype 3, 1 Year Post Vax 2 | 18 [14.2 to 22.3]
  Serotype 4, Pre Vax 2 | 710 [504.4 to 998.7]
  Serotype 4, 1 Year Post Vax 2 | 376 [264.2 to 534.0]
  Serotype 5, Pre Vax 2 | 39 [26.2 to 56.7]
  Serotype 5, 1 Year Post Vax 2 | 29 [20.4 to 42.1]
  Serotype 6A, Pre Vax 2 | 540 [347.1 to 838.8]
  Serotype 6A, 1 Year Post Vax 2 | 331 [227.1 to 483.3]
  Serotype 6B, Pre Vax 2 | 459 [292.2 to 719.9]
  Serotype 6B, 1 Year Post Vax 2 | 781 [529.8 to 1150.8]
  Serotype 7F, Pre Vax 2 | 146 [89.4 to 237.1]
  Serotype 7F, 1 Year Post Vax 2 | 244 [155.7 to 383.4]
  Serotype 9V, Pre Vax 2 | 96 [58.3 to 158.4]
  Serotype 9V, 1 Year Post Vax 2 | 201 [125.8 to 320.2]
  Serotype 14, Pre Vax 2 | 241 [159.6 to 364.0]
  Serotype 14, 1 Year Post Vax 2 | 383 [274.1 to 534.2]
  Serotype 18C, Pre Vax 2 | 403 [273.8 to 592.0]
  Serotype 18C, 1 Year Post Vax 2 | 398 [274.1 to 579.1]
  Serotype 19A, Pre Vax 2 | 203 [151.3 to 271.8]
  Serotype 19A, 1 Year Post Vax 2 | 253 [197.2 to 325.7]
  Serotype 19F, Pre Vax 2 | 114 [72.7 to 177.5]
  Serotype 19F, 1 Year Post Vax 2 | 238 [165.2 to 341.7]
  Serotype 23F, Pre Vax 2 | 90 [58.5 to 139.9]
  Serotype 23F, 1 Year Post Vax 2 | 104 [67.9 to 158.6]
Statistical Analysis 1: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; geometric mean fold rise = 1.0, 95% CI 2-sided [0.85 to 1.22] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; geometric mean fold rise = 1.0, 95% CI 2-sided [0.82 to 1.10] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; geometric mean fold rise = 0.5, 95% CI 2-sided [0.41 to 0.69] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; geometric mean fold rise = 0.8, 95% CI 2-sided [0.67 to 0.87] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; geometric mean fold rise = 0.6, 95% CI 2-sided [0.48 to 0.79] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; geometric mean fold rise = 1.7, 95% CI 2-sided [1.32 to 2.19] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); [analysis description as in outcome 4, analysis 19]; Test type: Superiority or Other; geometric mean fold rise = 1.7, 95% CI 2-sided [1.24 to 2.26] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; geometric mean fold rise = 2.1, 95% CI 2-sided [1.48 to 2.95] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); [analysis description as in outcome 4, analysis 25]; Test type: Superiority or Other; geometric mean fold rise = 1.6, 95% CI 2-sided [1.23 to 2.05] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); [analysis description as in outcome 4, analysis 28]; Test type: Superiority or Other; geometric mean fold rise = 1.0, 95% CI 2-sided [0.82 to 1.19] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); [analysis description as in outcome 4, analysis 31]; Test type: Superiority or Other; geometric mean fold rise = 1.2, 95% CI 2-sided [1.07 to 1.46] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); [analysis description as in outcome 4, analysis 34]; Test type: Superiority or Other; geometric mean fold rise = 2.1, 95% CI 2-sided [1.56 to 2.80] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC/13vPnC Group (23vPS Naïve); [analysis description as in outcome 4, analysis 37]; Test type: Superiority or Other; geometric mean fold rise = 1.1, 95% CI 2-sided [0.89 to 1.48] — [estimate comment as in outcome 2, analysis 1]

17. Secondary Outcome: Serotype-Specific Pneumococcal OPA GMT Antibody Persistence for 23vPS/13vPnC 1 Year After Vaccination 2 Compared to 13vPnC/13vPnC 1 Year After Vaccination 1 (Parent Study 6115A1-3005; NCT00546572)
Description: as for outcome 2
Time Frame: Month 0/Year 1 (Parent Study NCT00546572), Month 1/Year 2 (Baseline; Follow-up Study NCT01025336)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- 13vPnC (23vPS Vaccination ≥5 Years Prior): Participants at least 70 years of age or greater previously vaccinated with 23vPS ≥5 years before enrollment in the parent study 6115A1-3005 (NCT00546572), who completed study NCT00546572 receiving 13vPnC administered as a single dose 0.5 mL IM at Year 0 (Vaccination 1)
Arm/Group | 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior) | 13vPnC (23vPS Vaccination ≥5 Years Prior)
Number analyzed (Participants) | 222 | 220
titer
  Serotype 1 | 22 [17.5 to 27.8] | 33 [26.6 to 41.3]
  Serotype 3 | 16 [13.3 to 19.2] | 16 [13.5 to 19.6]
  Serotype 4 | 172 [129.0 to 230.1] | 123 [85.4 to 177.6]
  Serotype 5 | 42 [32.2 to 55.6] | 31 [24.4 to 40.2]
  Serotype 6A | 115 [84.5 to 156.8] | 271 [197.5 to 370.6]
  Serotype 6B | 381 [281.9 to 513.9] | 380 [274.0 to 526.3]
  Serotype 7F | 115 [81.6 to 160.9] | 61 [43.0 to 87.7]
  Serotype 9V | 68 [47.4 to 98.5] | 40 [27.8 to 58.3]
  Serotype 14 | 240 [181.0 to 317.0] | 126 [93.0 to 170.7]
  Serotype 18C | 360 [273.6 to 474.5] | 439 [343.4 to 559.9]
  Serotype 19A | 181 [146.7 to 222.9] | 183 [151.3 to 220.7]
  Serotype 19F | 158 [119.3 to 209.9] | 115 [87.4 to 151.3]
  Serotype 23F | 45 [33.5 to 59.6] | 59 [43.7 to 79.4]
Statistical Analysis 1: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 13vPnC (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; Ratio of GMT = 0.7, 95% CI 2-sided [0.48 to 0.92] — CIs for the ratio are back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures [(23vPS/13vPnC-13vPnC)]
Statistical Analysis 2: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 13vPnC (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; Ratio of GMT = 1.0, 95% CI 2-sided [0.76 to 1.28] — [estimate comment as in outcome 17, analysis 1]
Statistical Analysis 3: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 13vPnC (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 15, analysis 3]; Test type: Superiority or Other; Ratio of GMT = 1.4, 95% CI 2-sided [0.88 to 2.22] — [estimate comment as in outcome 17, analysis 1]
Statistical Analysis 4: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 13vPnC (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 15, analysis 4]; Test type: Superiority or Other; Ratio of GMT = 1.4, 95% CI 2-sided [0.93 to 1.95] — [estimate comment as in outcome 17, analysis 1]
Statistical Analysis 5: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 13vPnC (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; Ratio of GMT = 0.4, 95% CI 2-sided [0.27 to 0.66] — [estimate comment as in outcome 17, analysis 1]
Statistical Analysis 6: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 13vPnC (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 15, analysis 6]; Test type: Superiority or Other; Ratio of GMT = 1.0, 95% CI 2-sided [0.64 to 1.56] — [estimate comment as in outcome 17, analysis 1]
Statistical Analysis 7: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 13vPnC (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 15, analysis 7]; Test type: Superiority or Other; Ratio of GMT = 1.9, 95% CI 2-sided [1.14 to 3.04] — [estimate comment as in outcome 17, analysis 1]
Statistical Analysis 8: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 13vPnC (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 15, analysis 8]; Test type: Superiority or Other; Ratio of GMT = 1.7, 95% CI 2-sided [1.01 to 2.85] — [estimate comment as in outcome 17, analysis 1]
Statistical Analysis 9: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 13vPnC (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; Ratio of GMT = 1.9, 95% CI 2-sided [1.26 to 2.87] — [estimate comment as in outcome 17, analysis 1]
Statistical Analysis 10: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 13vPnC (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 15, analysis 10]; Test type: Superiority or Other; Ratio of GMT = 0.8, 95% CI 2-sided [0.57 to 1.19] — [estimate comment as in outcome 17, analysis 1]
Statistical Analysis 11: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 13vPnC (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 15, analysis 11]; Test type: Superiority or Other; Ratio of GMT = 1.0, 95% CI 2-sided [0.75 to 1.31] — [estimate comment as in outcome 17, analysis 1]
Statistical Analysis 12: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 13vPnC (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 15, analysis 12]; Test type: Superiority or Other; Ratio of GMT = 1.4, 95% CI 2-sided [0.93 to 2.04] — [estimate comment as in outcome 17, analysis 1]
Statistical Analysis 13: Comparison: 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 13vPnC (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 15, analysis 13]; Test type: Superiority or Other; Ratio of GMT = 0.8, 95% CI 2-sided [0.50 to 1.15] — [estimate comment as in outcome 17, analysis 1]

18. Secondary Outcome: Serotype-Specific Pneumococcal OPA GMT Antibody Persistence for 13vPnC/13vPnC 1 Year After Vaccination 2 Compared to 13vPnC/13vPnC After Vaccination 1 (Parent Study 6115A1-3005; NCT00546572)
Description: as for outcome 2
Time Frame: Month 0/Year 1 (Parent Study NCT00546572), Month 0/Year 2 (Baseline) (Follow-up Study 6115A1-3018; NCT01025336)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior)
Number analyzed (Participants) | 217
titer
  Serotype 1, Pre Vax 2 | 33 [26.4 to 41.1]
  Serotype 1, 1 Year Post Vax 2 | 38 [30.7 to 47.5]
  Serotype 3, Pre Vax 2 | 16 [13.2 to 19.4]
  Serotype 3, 1 Year Post Vax 2 | 19 [16.2 to 23.2]
  Serotype 4, Pre Vax 2 | 129 [89.0 to 186.9]
  Serotype 4, 1 Year Post Vax 2 | 267 [198.8 to 358.8]
  Serotype 5, Pre Vax 2 | 32 [25.0 to 41.4]
  Serotype 5, 1 Year Post Vax 2 | 57 [44.5 to 73.2]
  Serotype 6A, Pre Vax 2 | 279 [203.4 to 383.4]
  Serotype 6A, 1 Year Post Vax 2 | 256 [191.2 to 341.9]
  Serotype 6B, Pre Vax 2 | 403 [290.6 to 558.3]
  Serotype 6B, 1 Year Post Vax 2 | 511 [376.9 to 693.4]
  Serotype 7F, Pre Vax 2 | 66 [46.3 to 95.3]
  Serotype 7F, 1 Year Post Vax 2 | 175 [127.1 to 240.3]
  Serotype 9V, Pre Vax 2 | 40 [27.6 to 59.1]
  Serotype 9V, 1 Year Post Vax 2 | 76 [51.6 to 112.9]
  Serotype 14, Pre Vax 2 | 130 [96.1 to 176.2]
  Serotype 14, 1 Year Post Vax 2 | 204 [155.6 to 268.5]
  Serotype 18C, Pre Vax 2 | 436 [340.9 to 556.7]
  Serotype 18C, 1 Year Post Vax 2 | 545 [438.2 to 678.0]
  Serotype 19A, Pre Vax 2 | 185 [152.8 to 222.9]
  Serotype 19A, 1 Year Post Vax 2 | 235 [196.4 to 282.2]
  Serotype 19F, Pre Vax 2 | 121 [91.1 to 160.0]
  Serotype 19F, 1 Year Post Vax 2 | 261 [204.9 to 333.7]
  Serotype 23F, Pre Vax 2 | 60 [44.5 to 81.1]
  Serotype 23F, 1 Year Post Vax 2 | 104 [78.0 to 137.4]
Statistical Analysis 1: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; geometric mean fold rise = 1.2, 95% CI 2-sided [1.03 to 1.31] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; geometric mean fold rise = 1.2, 95% CI 2-sided [1.07 to 1.37] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; geometric mean fold rise = 2.1, 95% CI 2-sided [1.60 to 2.68] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 10]; Test type: Superiority or Other; geometric mean fold rise = 1.8, 95% CI 2-sided [1.55 to 2.03] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; geometric mean fold rise = 0.9, 95% CI 2-sided [0.79 to 1.07] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 16]; Test type: Superiority or Other; geometric mean fold rise = 1.3, 95% CI 2-sided [1.05 to 1.53] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 19]; Test type: Superiority or Other; geometric mean fold rise = 2.6, 95% CI 2-sided [1.98 to 3.50] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; geometric mean fold rise = 1.9, 95% CI 2-sided [1.37 to 2.61] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 25]; Test type: Superiority or Other; geometric mean fold rise = 1.6, 95% CI 2-sided [1.33 to 1.86] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 28]; Test type: Superiority or Other; geometric mean fold rise = 1.3, 95% CI 2-sided [1.10 to 1.42] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 31]; Test type: Superiority or Other; geometric mean fold rise = 1.3, 95% CI 2-sided [1.14 to 1.43] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 34]; Test type: Superiority or Other; geometric mean fold rise = 2.2, 95% CI 2-sided [1.80 to 2.60] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 4, analysis 37]; Test type: Superiority or Other; geometric mean fold rise = 1.7, 95% CI 2-sided [1.44 to 2.06] — [estimate comment as in outcome 2, analysis 1]

19. Secondary Outcome: Serotype-Specific Pneumococcal OPA GMT Antibody Persistence for 13vPnC 1 Year After Vaccination 1 Compared to 23vPS 1 Year After Vaccination 1 (Parent Study 6115A1-3010; NCT00574548)
Description: as for outcome 2
Time Frame: Month 0/Year 1 (Parent Study NCT00574548)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- 13vPnC (23vPS Naïve): Participants aged 60 to 64 years old who had never received 23vPS prior to enrollment into the parent study 6115A1-3010 (NCT00574548), completed study NCT00574548 receiving 13vPnC administered as a single dose 0.5 mL IM at Year 0 (Vaccination 1)
- 23vPS (23vPS Naïve): Participants aged 60 to 64 years old who had never been vaccinated with 23vPS prior to enrollment into the parent study (6115A1-3010 NCT00574548), who completed study NCT00574548 receiving 23vPS administered as a single dose 0.5 mL IM at Year 0 (Vaccination 1)
Arm/Group | 13vPnC (23vPS Naïve) | 23vPS (23vPS Naïve)
Number analyzed (Participants) | 332 | 175
titer
  Serotype 1 | 54 [45.4 to 65.0] | 45 [34.5 to 59.8]
  Serotype 3 | 21 [18.1 to 24.9] | 26 [20.4 to 32.5]
  Serotype 4 | 622 [496.9 to 777.7] | 332 [231.8 to 476.2]
  Serotype 5 | 52 [40.9 to 64.8] | 49 [36.4 to 66.9]
  Serotype 6A | 597 [466.8 to 764.7] | 82 [54.6 to 122.4]
  Serotype 6B | 420 [320.2 to 552.0] | 162 [108.9 to 241.6]
  Serotype 7F | 133 [99.6 to 177.8] | 66 [44.1 to 100.1]
  Serotype 9V | 85 [62.7 to 115.4] | 52 [33.7 to 80.3]
  Serotype 14 | 250 [193.5 to 324.2] | 302 [214.2 to 425.3]
  Serotype 18C | 439 [349.8 to 551.0] | 319 [222.5 to 457.3]
  Serotype 19A | 208 [175.9 to 245.7] | 153 [117.3 to 199.5]
  Serotype 19F | 147 [115.1 to 187.7] | 125 [88.8 to 176.5]
  Serotype 23F | 90 [69.9 to 116.6] | 30 [21.2 to 42.1]
Statistical Analysis 1: Comparison: 13vPnC (23vPS Naïve) vs 23vPS (23vPS Naïve); Serotype 1: Ratio of GMT (13vPnC to 23vPS) was calculated by back transforming the mean difference between vaccine group on the logarithmic scale; Test type: Superiority or Other; Ratio = 1.2, 95% CI 2-sided [0.87 to 1.64] — CIs for the GMFR are back transformations of a CI based on the Student t distribution for the mean logarithm of the measures [(13vPnC - 23vPS)]
Statistical Analysis 2: Comparison: 13vPnC (23vPS Naïve) vs 23vPS (23vPS Naïve); Serotype 3: Ratio of GMT (13vPnC to 23vPS) was calculated by back transforming the mean difference between vaccine group on the logarithmic scale; Test type: Superiority or Other; Ratio = 0.8, 95% CI 2-sided [0.63 to 1.08] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC (23vPS Naïve) vs 23vPS (23vPS Naïve); Serotype 4: Ratio of GMT (13vPnC to 23vPS) was calculated by back transforming the mean difference between vaccine group on the logarithmic scale; Test type: Superiority or Other; Ratio = 1.9, 95% CI 2-sided [1.25 to 2.80] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC (23vPS Naïve) vs 23vPS (23vPS Naïve); Serotype 5: Ratio of GMT (13vPnC to 23vPS) was calculated by back transforming the mean difference between vaccine group on the logarithmic scale; Test type: Superiority or Other; Ratio = 1.0, 95% CI 2-sided [0.71 to 1.53] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC (23vPS Naïve) vs 23vPS (23vPS Naïve); Serotype 6A: Ratio of GMT (13vPnC to 23vPS) was calculated by back transforming the mean difference between vaccine group on the logarithmic scale; Test type: Superiority or Other; Ratio = 7.3, 95% CI 2-sided [4.67 to 11.44] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 6: Comparison: 13vPnC (23vPS Naïve) vs 23vPS (23vPS Naïve); Serotype 6B: Ratio of GMT (13vPnC to 23vPS) was calculated by back transforming the mean difference between vaccine group on the logarithmic scale; Test type: Superiority or Other; Ratio = 2.6, 95% CI 2-sided [1.61 to 4.17] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC (23vPS Naïve) vs 23vPS (23vPS Naïve); Serotype 7F: Ratio of GMT (13vPnC to 23vPS) was calculated by back transforming the mean difference between vaccine group on the logarithmic scale; Test type: Superiority or Other; Ratio = 2.0, 95% CI 2-sided [1.22 to 3.29] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC (23vPS Naïve) vs 23vPS (23vPS Naïve); Serotype 9V: Ratio of GMT (13vPnC to 23vPS) was calculated by back transforming the mean difference between vaccine group on the logarithmic scale; Test type: Superiority or Other; Ratio = 1.6, 95% CI 2-sided [0.96 to 2.77] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC (23vPS Naïve) vs 23vPS (23vPS Naïve); Serotype 14: Ratio of GMT (13vPnC to 23vPS) was calculated by back transforming the mean difference between vaccine group on the logarithmic scale; Test type: Superiority or Other; Ratio = 0.8, 95% CI 2-sided [0.54 to 1.28] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC (23vPS Naïve) vs 23vPS (23vPS Naïve); Serotype 18C: Ratio of GMT (13vPnC to 23vPS) was calculated by back transforming the mean difference between vaccine group on the logarithmic scale; Test type: Superiority or Other; Ratio = 1.4, 95% CI 2-sided [0.92 to 2.07] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC (23vPS Naïve) vs 23vPS (23vPS Naïve); Serotype 19A: Ratio of GMT (13vPnC to 23vPS) was calculated by back transforming the mean difference between vaccine group on the logarithmic scale; Test type: Superiority or Other; Ratio = 1.4, 95% CI 2-sided [1.01 to 1.83] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 12: Comparison: 13vPnC (23vPS Naïve) vs 23vPS (23vPS Naïve); Serotype 19F: Ratio of GMT (13vPnC to 23vPS) was calculated by back transforming the mean difference between vaccine group on the logarithmic scale; Test type: Superiority or Other; Ratio = 1.2, 95% CI 2-sided [0.77 to 1.78] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC (23vPS Naïve) vs 23vPS (23vPS Naïve); Serotype 23F: Ratio of GMT (13vPnC to 23vPS) was calculated by back transforming the mean difference between vaccine group on the logarithmic scale; Test type: Superiority or Other; Ratio = 3.0, 95% CI 2-sided [1.97 to 4.64] — [estimate comment as in outcome 19, analysis 1]

20. Secondary Outcome: Serotype-Specific Pneumococcal OPA GMT Antibody Persistence for 13vPnC 1 Year After Vaccination 1 Compared to 23vPS 1 Year After Vaccination 1 (Parent Study 6115A1-3005; NCT00546572)
Description: as for outcome 2
Time Frame: Month 0/Year 1 (Parent Study NCT00546572)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) | 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior)
Number analyzed (Participants) | 220 | 222
titer
  Serotype 1 | 33 [26.6 to 41.3] | 21 [16.8 to 26.5]
  Serotype 3 | 16 [13.5 to 19.6] | 16 [13.2 to 19.8]
  Serotype 4 | 123 [85.4 to 177.6] | 68 [47.0 to 96.9]
  Serotype 5 | 31 [24.4 to 40.2] | 23 [17.6 to 29.7]
  Serotype 6A | 271 [197.5 to 370.6] | 57 [40.9 to 78.2]
  Serotype 6B | 380 [274.0 to 526.3] | 168 [118.6 to 238.1]
  Serotype 7F | 61 [43.0 to 87.7] | 63 [43.8 to 91.1]
  Serotype 9V | 40 [27.8 to 58.3] | 29 [20.3 to 41.3]
  Serotype 14 | 126 [93.0 to 170.7] | 140 [101.7 to 192.7]
  Serotype 18C | 439 [343.4 to 559.9] | 271 [197.8 to 371.7]
  Serotype 19A | 183 [151.3 to 220.7] | 122 [96.0 to 155.9]
  Serotype 19F | 115 [87.4 to 151.3] | 86 [63.2 to 115.9]
  Serotype 23F | 59 [43.7 to 79.4] | 30 [22.3 to 41.0]
Statistical Analysis 1: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; Ratio = 1.6, 95% CI 2-sided [1.15 to 2.15] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 2: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 19, analysis 2]; Test type: Superiority or Other; Ratio = 1.0, 95% CI 2-sided [0.76 to 1.32] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 19, analysis 3]; Test type: Superiority or Other; Ratio = 1.8, 95% CI 2-sided [1.09 to 3.05] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 19, analysis 4]; Test type: Superiority or Other; Ratio = 1.4, 95% CI 2-sided [0.95 to 1.96] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 19, analysis 5]; Test type: Superiority or Other; Ratio = 4.8, 95% CI 2-sided [3.05 to 7.50] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 6: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 19, analysis 6]; Test type: Superiority or Other; Ratio = 2.3, 95% CI 2-sided [1.40 to 3.64] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 19, analysis 7]; Test type: Superiority or Other; Ratio = 1.0, 95% CI 2-sided [0.58 to 1.62] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 19, analysis 8]; Test type: Superiority or Other; Ratio = 1.4, 95% CI 2-sided [0.83 to 2.32] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 19, analysis 9]; Test type: Superiority or Other; Ratio = 0.9, 95% CI 2-sided [0.58 to 1.40] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 19, analysis 10]; Test type: Superiority or Other; Ratio = 1.6, 95% CI 2-sided [1.09 to 2.41] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 19, analysis 11]; Test type: Superiority or Other; Ratio = 1.5, 95% CI 2-sided [1.10 to 2.03] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 12: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 19, analysis 12]; Test type: Superiority or Other; Ratio = 1.3, 95% CI 2-sided [0.89 to 2.02] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) vs 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior); [analysis description as in outcome 19, analysis 13]; Test type: Superiority or Other; Ratio = 1.9, 95% CI 2-sided [1.27 to 2.97] — [estimate comment as in outcome 19, analysis 1]

21. Primary Outcome: Serotype-Specific Pneumococcal OPA GMT Antibody Persistence 1 Year After Vaccination 2 in Parent Study 6115A1-3005 (NCT00546572)
Description: as for outcome 1
Time Frame: Month 1/Year 2 (Baseline) (Follow-up Study 6115A1-3018; NCT01025336)
Population: All-Available Immunogenicity Population. N=number of participants with valid and determinate antibody titer for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) | 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior)
Number analyzed (Participants) | 220 | 222
titer
  Serotype 1 | 38 [30.9 to 47.9] | 22 [17.5 to 27.8]
  Serotype 3 | 20 [16.5 to 23.4] | 16 [13.3 to 19.2]
  Serotype 4 | 265 [200.8 to 348.5] | 172 [129.0 to 230.1]
  Serotype 5 | 58 [45.1 to 74.1] | 42 [32.2 to 55.6]
  Serotype 6A | 250 [187.3 to 334.0] | 115 [84.5 to 156.8]
  Serotype 6B | 510 [378.2 to 686.4] | 381 [281.9 to 513.9]
  Serotype 7F | 173 [126.0 to 237.5] | 115 [81.6 to 160.9]
  Serotype 9V | 81 [55.1 to 117.9] | 68 [47.4 to 98.5]
  Serotype 14 | 202 [154.6 to 265.0] | 240 [181.0 to 317.0]
  Serotype 18C | 540 [435.5 to 668.5] | 360 [273.6 to 474.5]
  Serotype 19A | 232 [193.2 to 278.1] | 181 [146.7 to 222.9]
  Serotype 19F | 277 [218.6 to 351.7] | 158 [119.3 to 209.9]
  Serotype 23F | 103 [78.0 to 135.5] | 45 [33.5 to 59.6]

ADVERSE EVENTS:
Arm/Group | 13vPnC/13vPnC Group (23vPS Naïve) | 13vPnC/23vPS Group (23vPS Naïve) | 23vPS/13vPnC Group (23vPS Naïve) | 13vPnC/13vPnC Group (23vPS Vaccination ≥5 Years Prior) | 23vPS/13vPnC Group (23vPS Vaccination ≥5 Years Prior)
Serious Adverse Events (participants affected / at risk) | 0/130 | 0/210 | 0/179 | 0/221 | 0/222
Other Adverse Events (participants affected / at risk) | 0/130 | 0/210 | 0/179 | 0/221 | 0/222

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.